## **CONVOCATORIA 841 DE COLCIENCIAS**

**TÍTULO DEL PROYECTO:** Rediseño, implementación y evaluación de la efectividad de la prótesis mioeléctrica Aktio

## **INVESTIGADOR PRINCIPAL Y COINVESTIGADORES**

Jenny Kateryne Aristizabal Nieto (Investigadora principal)

Juan Diego Lemos Duque (Coinvestigador)

Juan Guillermo Barreneche (Coinvestigador)

Sofía Catalina Henao Aguirre (Coinvestigadora)

Ana María Posada (Coinvestigadora)

Sara Salazar Salgado (Coinvestigadora)

Estefanía Aramburo (Coinvestigadora)

Jorge Robledo (Coinvestigador)

Juan Gabriel Arboleda (Coinvestigador)

Luis Horacio Atehortúa López (Coinvestigador)

Meisser Alberto López Córdoba (Coinvestigador)

Juan Carlos Parra Peláez (Coinvestigador)

Luz Ángela Calderón Calderón (Coinvestigadora)

# CONFORMACIÓN DEL EQUIPO DE INVESTIGACIÓN

| Nombre | Jenny Kateryne Aristizabal Nieto |
|---|---|
| Identificación | 1.128.267.261 |
| Institución | Universidad de Antioquia. Grupo de Investigación en Bioinstrumentación e Ingeniería Clínica (GIBIC) - COL0054963 |
| Funciones | Liderar el proyecto, verificar el diseño experimental y metodológico, liderar el diseño y fabricación de la prótesis. Participar en la escritura y revisión de artículos científicos y comunicaciones a congresos. Velar por la ejecución del proyecto de acuerdo con lo previsto. |
| Dedicación | 10 horas/semana, 36 meses |

| Nombre | Juan Diego Lemos Duque |
|---|---|
| Identificación | 71.774.114 |
| Institución | Universidad de Antioquia. Grupo de Investigación en Bioinstrumentación e Ingeniería Clínica (GIBIC) - COL0054963 |
| Funciones | Liderar el diseño electrónico y fabricación de la prótesis. Participar en la escritura y revisión de artículos científicos y comunicaciones a congresos. |

| Dedicación | 2 horas/semana, 36 meses |
|---|---|
| Nombre | Juan Guillermo Barreneche |
| Identificación | 8.129.113 |
| Institución | Universidad de Antioquia. Grupo de Investigación en Bioinstrumentación e Ingeniería Clínica (GIBIC) - COL0054963 |
| Funciones | Liderar la evaluación financiera, económica y comercial de la prótesis. Participar en la escritura y revisión de artículos científicos y comunicaciones a congresos. |
| Dedicación | 5 horas/semana, 36 meses |
| Nombre | Sofía Catalina Henao Aguirre |
| Identificación | 32.259.884 |
| Institución | Universidad de Antioquia. Grupo de Investigación en Bioinstrumentación e Ingeniería Clínica (GIBIC) - COL0054963 |
| Funciones | Liderar el diseño mecánico y fabricación de la prótesis. Participar en la escritura y revisión de artículos científicos y comunicaciones a congresos. |
| Dedicación | 5 horas/semana, 36 meses |
| Namahan | AINI |
| Nombre | NN |
| Identificación | NN |
| Institución | Universidad de Antioquia. Grupo de Investigación en Bioinstrumentación e Ingeniería Clínica (GIBIC) - COL0054963 |
| Funciones | Estudiante de maestría encargado del diseño mecánico de la prótesis. Analizar los resultados del estudio de efectividad. Escribir artículos científicos y participar en congresos. |
| Dedicación | 40 horas/semana, 24 meses |
| Nombre | Ana María Posada Borrero |
| Identificación | 43.272.550 |
| Institución | Universidad de Antioquia. Grupo de Investigación Rehabilitación en Salud - COL0015599 |

| Funciones | Verificar el cumplimiento de los aspectos metodológicos del estudio de efectividad, los criterios de inclusión y exclusión y la aleatorización de la intervención. Participar en la escritura y revisión de artículos científicos y comunicaciones a congresos y en las funciones asignadas por el investigador principal. |
|---|---|
| Dedicación | 4 horas/semana, 36 meses |

| Nombre | Sara Salazar Salgado |
|---|---|
| Identificación | 1.128.279.803 |
| Institución | Prótesis Avanzadas S.A.S. |
| Funciones | Asesorar y participar en la fase de diseño conceptual en la obtención de información de los usuarios y el staff médico. Acompañar en la búsqueda bibliográfica a lo largo del proyecto. Participar en la generación de ideas y fabricación de los prototipos a probar en los usuarios. Participar en el análisis de resultados del estudio de efectividad. Participar en la escritura y revisión de artículos científicos y comunicaciones a congresos y en las funciones asignadas por el investigador principal. |
| Dedicación | 10 horas/semana, 36 meses |

| Nombre | Estefanía Aramburo |
|---|---|
| Identificación | 1.017.219.914 |
| Institución | Prótesis Avanzadas S.A.S. |
| Funciones | Acompañar en el proceso de diseño y fabricación de la nueva prótesis. Participar en la escritura y revisión de artículos científicos y comunicaciones a congresos y en las funciones asignadas por el investigador principal. |
| Dedicación | 10 horas/semana, 36 meses |

| Nombre | Jorge Robledo |
|---|---|
| Identificación | 3.396.483 |
| Institución | Prótesis Avanzadas S.A.S. |
| Funciones | Acompañar en el proceso de diseño y fabricación de la prótesis mioeléctrica, asesorando en las áreas de mecánica, electrónica, sensores mioeléctricos, diseño CAD e impresión 3D |

| Dedicación | 10 horas/semana, 36 meses |
|---|---|
| Nombre | Juan Gabriel Arboleda |
| Identificación | 1.037.603.621 |
| Institución | Prótesis Avanzadas S.A.S. |
| Funciones | Liderar la evaluación financiera, económica y comercial de la prótesis. Participar en la escritura y revisión de artículos científicos y comunicaciones a congresos. |
| Dedicación | 10 horas/semana, 36 meses |
| Nombre | Luis Horacio Atehortúa López |
| I dan Miliana ai dan | 70.454.000 |

| Nombre | Luis Horacio Atehortúa López |
|---|---|
| Identificación | 79.154.292 |
| Institución | Fundación Hospitalaria San Vicente de Paúl. Investigación Clínica Aplicada - COL0171235 |
| Funciones | Internista, Intensivista y Magíster en Gestión de CTel, que asesorará el diseño y evaluación de la nueva prótesis, además de apoyar las labores de gestión del proyecto dentro de la Fundación Hospitalaria San Vicente de Paúl. |
| Dedicación | 2 horas/semana, 36 meses |

| Nombre | Meisser Alberto López Córdoba |
|---|---|
| Identificación | 73.143.394 |
| Institución | Fundación Hospitalaria San Vicente de Paúl. Investigación Clínica Aplicada - COL0171235 |
| Funciones | Médico especialista en Ortopedia y Cirujano de Mano que asesorará el diseño y evaluación de la nueva prótesis desde la perspectiva de su especialidad médica. |
| Dedicación | 2 horas/semana, 36 meses |

| Nombre | Juan Carlos Parra Peláez |
|---|---|
| Identificación | 15.384.135 |
| Institución | Fundación Hospitalaria San Vicente de Paúl. Investigación Clínica Aplicada - COL0171235 |

| Funciones | Médico especialista en Fisiatría y Rehabilitación que asesorará el diseño y evaluación de la nueva prótesis desde la perspectiva de su especialidad médica. |
|---|---|
| Dedicación | 2 horas/semana, 36 meses |

| Nombre | Luz Ángela Calderón |
|---|---|
| Identificación | 1.102.361.066 |
| Institución | Fundación Hospitalaria San Vicente de Paúl. Investigación Clínica Aplicada - COL0171235 |
| Funciones | Terapeuta ocupacional encargada del entrenamiento de pacientes en el uso de la prótesis, y de la realización de las pruebas para la evaluación de efectividad. Además, hará parte de los grupos focales de la fase de diseño. |
| Dedicación | 10 horas/semana, 12 meses |

| Nombre | NN |
|---|---|
| Identificación | NA |
| Institución | NA |
| Funciones | Ingeniero encargado del diseño electrónico de la prótesis. Analizar los resultados del estudio de efectividad. Escribir artículos científicos y participar en congresos. |
| Dedicación | 20 horas/semana, 12 meses |

# TRAYECTORIA DEL EQUIPO DE INVESTIGACIÓN

Las instituciones proponentes del presente proyecto tienen experiencia desarrollando proyectos de innovación e investigación relacionados con la biomecánica y la rehabilitación de personas en situación de discapacidad.

A continuación, se describen los grupos de investigación e instituciones que conforman el equipo que presenta esta propuesta.

UNIVERSIDAD DE ANTIOQUIA: Grupo de Investigación en Bioinstrumentación e Ingeniería Clínica (GIBIC). Código GrupLac: COL0054963

Líder: Mauricio Hernández Categoría Colciencias: B El grupo de Investigación en Bioinstrumentación e Ingeniería Clínica (GIBIC) es un grupo asociado al programa de Bioingeniería de la Universidad de Antioquia. Su campo de investigación es la Ingeniería Biomédica, campo desde el cual ha liderado proyectos de investigación aplicada, y de investigación y desarrollo. Una de sus líneas de investigación se centra en la biomecánica y rehabilitación física, y en dicha línea se han realizado las siguiente publicaciones:

- 1. Parametric Modeling of Kinetic-Kinematic Polycentric Mechanical Knee. In: VII Latin American Congress on Biomedical Engineering CLAIB 2016, Bucaramanga, Santander, Colombia, October 26th -28th, 2016. IFMBE Proceedings, vol 60. Springer, Singapore.
- 2. Classification Techniques for the Recognition of Neuromuscular Diseases. In: Memorias Congreso Iberoamericano de Tecnologías de Apoyo a la Discapacidad, Bogotá, Cundinamerca, Colombia. ISBN: 2619-6433, p.68 75, 2017.
- 3. Gait Parameters Identification for Differentiation of Neurodegenerative Diseases using Classifiers, 2017 Global Medical Engineering Physics Exchanges/Pan American Health Care Exchanges (GMEPE/PAHCE), Tuxtla Gutierrez, 2017, pp. 1-3. doi: 10.1109/GMEPEPAHCE.2017.7972076.
- 4. Design and Validation of an Alignment Protocol for Mechanical Prostheses Based on a Multivariate Biomechanical Model", Memorias Congreso Iberoamericano de Tecnologías de Apoyo a la Discapacidad IBERDISCAP 2017.

De igual manera, el grupo de investigación cuenta 4 trabajos de grado en estos mismos temas:

- 1. Desarrollo de un módulo de entrenamiento en cirugía de columna implementado en la plataforma Daubara (2016).
- Evaluación de los efectos de una implantación quirúrgica imprecisa en prótesis de cadera tipo resurfacing por medio de elementos finitos, con el fin de prevenir el fallo prematuro - (2017).
- Identificación de las variables cinéticas, cinemáticas y funcionales en el proceso de adaptación protésica y la rehabilitación postprotésica en pacientes amputados de miembro inferior - (2018).
- 4. Diseño de un juego serio orientado a la rehabilitación con prótesis de miembro inferior (2018).

Actualmente, el grupo de investigación tiene 1 estudiante de maestría y 1 estudiante de doctorado activos, cuyos trabajos incluyen también temas en el área de biomecánica y rehabilitación:

- 1. Tesis de maestría en curso. Dispositivo de alineación para prótesis transfemorales.
- Tesis de doctorado en curso. Diseño y validación de un protocolo de alineación de prótesis mecánicas con rodilla poliaxial, basado en un modelo biomecánico multivariado.

Así mismo, el grupo de investigación GIBIC cuenta con experiencia en la ejecución de un proyecto de investigación financiado por Colciencias con código de registro 63475 en la convocatoria 808-2018 "Contribución a los retos de país" en la línea temática "Soluciones contra minas antipersonales y artefactos improvisados" relacionado con el diseño de un estrategia combinada para mejorar la adherencia de sujetos amputados por artefactos explosivos improvisados al uso de prótesis de miembro inferior.

# UNIVERSIDAD DE ANTIOQUIA: Grupo de Investigación Rehabilitación en Salud. Código GrupLac: COL0015599

Líder: Luz Helena Lugo Agudelo

Categoría Colciencias: A

# Líneas de investigación

- 1. Funcionamiento y rehabilitación en adultos: Electrodiagnóstico, lesión medular, rehabilitación cardiaca y ejercicio terapéutico y accidentes de tránsito.
- 2. Funcionamiento y rehabilitación en niños: Calidad de vida, discapacidad intelectual.
- 3. Investigación en tecnologías en Rehabilitación.
- 4. Validación de escalas de funcionamiento, calidad de vida y participación.
- 5. Traslación del conocimiento en rehabilitación. Elaboración e implementación de guías de práctica clínica.

# Proyectos activos

- 1. Identificación de facilitadores y barreras para la implementación de la Guía de Práctica Clínica de diagnóstico y tratamiento preoperatorio, intraoperatorio y postoperatorio de la persona amputada, la prescripción de la prótesis y la rehabilitación integral.
- 2. Modelo para el desarrollo humano y ocupacional de personas con discapacidad intelectual. Métodos mixtos.
- 3. Efectividad de una estrategia basada en Telesalud para mejorar la implementación de la Guía de Práctica Clínica para el diagnóstico y tratamiento preoperatorio, intraoperatorio y postoperatorio de la persona amputada, la prescripción de la prótesis y la rehabilitación integral en instituciones de salud en Antioquia: Un estudio de intervención aleatorizado por conglomerados de hospitales.
- 4. Factores asociados al reintegro ocupacional un año después en pacientes con trauma craneoencefálico moderado y grave ocurrido en Medellín y su área metropolitana entre 2018 y 2019. Estudio de cohorte.
- 5. Efectividad de un programa de rehabilitación cardiaca fase III en pacientes con falla cardíaca.

#### Publicaciones relacionadas

- López-Posada J, Plata-Contreras J, Lugo-Agudelo L. Evaluación de la calidad de guías de práctica clínica en personas que han sufrido amputación de miembro inferior: revisión de la literatura y evaluación con el instrumento AGREE II. IATREIA 2016; 29(4-S2): S59-71.
- 2. Posada-Borrero A, Plata-Contreras J, Lugo-Agudelo L. Participación de los pacientes con amputación del miembro inferior en la elaboración de una guía de práctica clínica en Colombia. IATREIA 2016; 29(4-S2): S96-109.
- Puerta-Gómez A, Lugo-Agudelo L, Castaño-González A, Posada-Borrero A, López-Posada J, Valderrama-Molina C. Reconstrucción versus amputación en pacientes con lesiones graves del miembro inferior. Recomendaciones basadas en la evidencia para la Guía de Práctica Clínica de personas amputadas de miembro inferior en Colombia. IATREIA 2016; 29(4-S2):S72-81.
- 4. Salinas-Durán F, Ahunca L, Muñoz-Rodríguez D, Vélez-Jaramillo D, Sierra Abaunza J, Lugo-Agudelo L. Guía de práctica clínica para el diagnóstico y tratamiento preoperatorio, intraoperatorio y postoperatorio de la persona amputada, la

- prescripción de la prótesis y la rehabilitación integral Recomendaciones para el Tratamiento de Rehabilitación en adultos amputados. IATREIA 2016; 29(4-S2):S96-109.
- 5. Castaño-González A, Ceballos-González M, Vera-Giraldo C, Lugo-Agudelo I. Funcionamiento y estado de salud en una población de amputados de miembro inferior en Medellín, Colombia. IATREIA 2016; 29(4-S2):S122-135.
- Ceballos M, Orozco L, Valderrama C, Londoño D, Lugo L. Cost-Effectiveness Analysis
  of the Use of a Prophylactic Antibiotic for Patients Undergoing Lower Limb Amputation
  due to Diabetes or Vascular Illness in Colombia. Ann. vasc. surg. 2017;40:327-334.
  doi: 10.1016/j.avsg.2016.07.090.
- 7. Ceballos M, Valderrama C, Orozco L, Sánchez L, Valderrama JP, Lugo LH. Cost-Utility Analysis of Reconstruction Compared With Primary Amputation for Patients With Severe Lower Limb Trauma in Colombia. J Orthop Trauma. 2017;24(9):e288-e294.

# FUNDACIÓN HOSPITALARIA SAN VICENTE DE PAUL: Investigación Clínica Aplicada - COL0171235

Líder: Fabián Alberto Jaimes Barragán

Categoría Colciencias: C

## Líneas de investigación

- 1. Calidad y cuidado de enfermería
- 2. Endocrinología
- 3. Hospital rehabilitador
- 4. Infectología y microbiología
- 5. Informática en ciencias de la salud y el bienestar humano
- 6. Ingeniería y desarrollo aplicados a la salud
- 7. Investigación cardiovascular (GICARDIO)
- 8. Laboratorio de investigación en psiquiatría de enlace y medicina psicosomática
- 9. Morbilidad y mortalidad hospitalaria
- 10. Médicina de laboratorio
- 11. Neuroestimulación
- 12. Oncología
- 13. Reumatología
- 14. Vigilancia Farmacológica

## Proyectos activos

- Estudio piloto aleatorizado como prueba de concepto de cirugía coronaria con inyección de WJ-MSC y colocación de un parche epicárdico de matriz extracelular sembrado con WJ-MSC en pacientes con cardiomiopatía isquémica.
- 2. Mecanismos de daño y disfunción endotelial en el síndrome antifosfolípido. ¿hay diferencias de acuerdo a las manifestaciones clínicas del sindrome?
- 3. Determinación del balance activación/regulación del complemento en los transtornos hipertensivos en Colombia.
- Costo-Efectividad del tratamiento intrahospitalario de úlceras por presión en pacientes hospitalizados entre el periodo 2005-2016. Hospital Universitario San Vicente Fundación.

- 5. Determinar la presencia de interferencia en el registro del EEG y EKG, en pacientes con Dispositivos de Estimulación Cerebral Profunda implantados en Centros Especializados de San Vicente Fundación de Rionegro.
- 6. Estabilidad de los parámetros del citoquimico del líquido cefalorraquídeo en diferentes tiempos y condiciones de almacenamiento.
- 7. Identificación de microorganismos en bilis de pacientes cirroticos en el momento del trasplante hepatico. rompiendo paradigmas.
- 8. Conocimientos, actitudes y prácticas sobre la donación de órganos en diferentes poblaciones en Antioquia.
- 9. Niveles de glucemia intraoperatoria y su relación con resultados a corto y largo plazo en pacientes trasplantados de hígado.
- 10. Estudio para validación de tecnología de dispositivo medico: Neumobarometro digital desarrollado por el área de ingeniería biomédica de HUSVF.
- 11. Supervivencia de los pacientes con enfermedad renal cronica terminal segun el periodo de ingreso al programa de hemodialisis entre 1981 y 2014.
- 12. Terapia transfusional preoperatoria e intraoperatoria guiada por Tromboelastografía y pruebas de coagulación convencional en pacientes sometidos a trasplante hepático, San Vicente Fundación: Estudio observacional retrospectivo.
- 13. Características clínicas y supervivencia libre de enucleación en pacientes con retinoblastoma tratados con quimioterapia intraarterial atendidos en el Hospital Universitario San Vicente Fundación.
- 14. Infección por VIH sida en unidad de cuidados intensivos: Descripción del perfil epidemiológico de una cohorte multicéntrica local.
- 15. Complicaciones vasculares en pacientes trasplantados hepáticos en el Hospital San Vicente Fundación.
- 16. Factores de riesgo asociados a enfermedad tromboembolica venosa en un hospital de alta complejidad.

# Publicaciones relacionadas

- 1. Ronda clínica y epidemiológica. Series de tiempo interrumpidas.
- Factores asociados a la percepción del estado de salud en habitantes de calle de Medellín.

# Prótesis Avanzadas S.A.S.

La empresa Prótesis Avanzadas S.A.S. se ha dedicado, desde hace casi 4 años, al diseño, fabricación y comercialización de prótesis mioeléctricas de miembro superior a nivel transradial (*i.e.* debajo de codo). Integrando funcionalidad, tecnología y estética, ofrece un producto fabricado en impresión 3D, de bajo costo, que permite realizar actividades de la vida cotidiana, y por lo tanto, recuperar la independencia de sus usuarios. Desde el año 2016, cuenta con el certificado de condiciones sanitarias y el registro sanitario para la fabricación y venta del dispositivo médico mano robótica con control mioeléctrico. En el mismo año, obtuvo la patente de modelo de utilidad de la prótesis mioeléctrica de mano obtenida por impresión 3D con movimiento mejorado del pulgar y en el año 2018 se certificó para la elaboración y adaptación de dispositivos médicos sobre medida de tecnología ortopédica externa, correspondiente a la prótesis mioeléctrica transradial. Actualmente cuenta con 37 prótesis adaptadas, 34 de ellas a nivel nacional y 3 en el exterior.

# TEMÁTICA DE INVESTIGACIÓN

Este proyecto se enmarca en la temática de "Discapacidad, habilitación y rehabilitación e incidente vial", la cual se enfoca en dispositivos médicos, implantes quirúrgicos, tejidos artificiales y prótesis.

#### **RESUMEN EJECUTIVO**

En Latinoamérica, Colombia ocupa el cuarto lugar en países con mayores cifras de personas con discapacidad (6,4%), el 80% de estos vive en estratos 1 y 2, tienen poco acceso a la educación y altas tasas de desempleo. De estos casi 3 millones de personas con esta condición, se estima que 11.476 necesitan prótesis de miembro superior, 12% de las cuales tienen amputación transradial o por encima del codo. A pesar de que muchas de las funciones que se han perdido por la amputación pueden recuperarse con una prótesis, en Colombia pocas personas usan estos dispositivos. Esto se debe a que, actualmente, solo se encuentran opciones estéticas y mecánicas, y las opciones más avanzadas como las mioeléctricas, son fabricadas en otros países tienen precios muy elevados y no están diseñadas según las necesidades locales. La única opción fabricada a nivel nacional es la desarrollada por Prótesis Avanzadas S.A.S., pero que todavía tiene aspectos a mejorar que la llevarían a adaptarse de una mejor manera a las necesidades de los usuarios colombianos.

Todo lo anterior muestra la evidente necesidad que tiene el país de generar productos que puedan ayudar a esta población. El objetivo de este proyecto es entonces rediseñar, implementar y evaluar la efectividad de una prótesis mioeléctricas transradial de buena calidad, enfocadas en la población amputada colombiana y que mejoren los índices de aceptación. Para la fase de diseño del estudio se incluirá un grupo conformado por profesionales de la salud y pacientes con amputación transradial para evaluar las preferencias y prioridades de su prótesis. Para la validación pre-comercial, se realizará un estudio de efectividad mediante un ensayo clínico cruzado aleatorizado con 12 participantes en los que se analizará el funcionamiento y la calidad de vida del usuario con y sin la prótesis y la satisfacción con la misma usando métodos de estimación bayesianos. Con este estudio se espera no solo mejorar la calidad de vida de las personas con amputación transradial y de sus familias, sino también brindar una opción funcional para las ARL y el sistema de salud.

## **PALABRAS CLAVES**

Prótesis de miembro superior, prótesis mioeléctrica, transradial, impresión 3D, adherencia.

# JUSTIFICACIÓN DEL PROYECTO

Según el Banco Mundial y la Organización Mundial de la Salud (OMS), aproximadamente 1.000 millones de personas tienen algún tipo de discapacidad, lo que la convierte en la mayor minoría del mundo [1], [2]. Según el programa de las Naciones Unidas para el Desarrollo (PNUD), aproximadamente el 80% de esta población vive en países en vía de desarrollo con bajos ingresos económicos. Según la Organización Internacional del Trabajo (OIT), 386 millones de personas que integran el grupo de personas con discapacidad están en edad de trabajar; sin embargo, la mayoría de ellos son desempleados, alcanzando tasas de desempleo en algunos países de hasta 80%. En Estados Unidos, por ejemplo, la tasa de desempleo para personas con discapacidad es de aproximadamente 65%, mientras que la

de personas sin esta condición es del 22%. La mayoría de los desempleados con discapacidad expresaron que les gustaría trabajar, pero no les era posible encontrar un empleo, probablemente por no contar con las condiciones adecuadas para desempeñarlo [3].

Según registros que comparan los censos nacionales de varios países de latinoamérica, Colombia ocupa el cuarto lugar en mayores cifras de personas en situación de discapacidad (6,4%); luego de Brasil (14,9%), Perú (10,9%) y Argentina (7,1%) [4]. De estos casi tres millones de colombianos, el 49% vive en estrato 1, el 33% en estrato 2 y el 14% en estrato 3. En cuanto al tema de ingresos, el 64,12% no cuenta con ningún ingreso y el 21,33% vive con menos de \$500.000 al mes, lo que suma más del 80% de la población con esta condición. En cuanto al trabajo, según el Registro de Localización y Caracterización de Personas con Discapacidad (RLCPD), en Colombia, el 32% de esta población no cuenta con pensión y está incapacitado permanentemente para trabajar, el 18% realiza trabajos del hogar y solo el 12% cuenta con un trabajo [5].

Específicamente, hablando de amputaciones, se estima que en el mundo habitan aproximadamente 40 millones de amputados; no obstante, debido en parte al envejecimiento de la población, se cree que este número será aproximadamente el doble en el año 2050 [6]. De estos 40 millones de amputados, aproximadamente el 3% corresponde a amputaciones de miembro superior [7]. A pesar de la diferencia, la pérdida de la extremidad superior altera de forma más significativa la vida de una persona debido a la complejidad de la anatomía de la mano y a las múltiples funciones que esta realiza [8]–[11].

En Colombia, según cifras del DANE, casi un 40% de las personas con discapacidad presentan limitaciones en el movimiento del cuerpo, manos, brazos y piernas; grupo donde se incluirían las amputaciones o pérdida de alguna(s) extremidad(es) [5], [12]. Aunque no se cuenta con una cifra exacta de esta condición, según datos del Cubo de Discapacidad del Sistema Integral de Información de la Protección Social, del 28 de mayo de 2018, se reportan 11.476 personas que necesitan prótesis de miembro superior [13].

Las causas de amputación de miembros superiores van desde trauma (accidentes laborales o de tránsito), hasta cáncer, problemas vasculares y deficiencias congénitas [14]. Estas amputaciones incluyen pérdida del brazo y partes del tronco (inter-toraco-escapular), de todo el brazo (desarticulado de hombro), partes de este (transhumeral o transradial) o la mano o partes de ella (desarticulado de muñeca o amputaciones parciales) [9], [11], [15]. De estos, el porcentaje de amputaciones parciales de mano es del 61%, mientras que las transhumerales corresponden al 16%, las transradiales al 12%, y las demás tienen valores menores al 3% cada una [9].

Para las personas que han sufrido de una amputación de miembro superior, parte de su rehabilitación es contar con una prótesis que les permita recuperar en cierta forma la función perdida, permitiéndoles ganar autonomía y mejorar su calidad de vida. Según el RLCPD, el 80% de las personas en situación de discapacidad tienen acceso a la rehabilitación a través del sistema general de salud, el cual, según la ley, está obligado a proporcionar prótesis para las personas amputadas [5]. Con respecto a las leyes colombianas, en la Ley 1751 de 2015 se regula el derecho fundamental a la salud incluyendo, entre otros, la provisión y acceso oportuno a las tecnologías y a los medicamentos requeridos, así como a agotar las posibilidades de tratamiento para la superación de la enfermedad [16]. Así mismo, el

Congreso de Colombia determina las disposiciones para garantizar el pleno ejercicio de los derechos de las personas con discapacidad y establece mecanismos para su integración social, por medio de la Ley 1618 y la Ley 361, respectivamente, otorgando la facultad de acceder a los procesos de habilitación y rehabilitación integral con el objetivo de lograr y mantener la máxima autonomía e independencia, en su capacidad física, mental y vocacional, así como la inclusión y participación plena en todos los aspectos de la vida [17]. Además, dicta que los municipios podrán destinar recursos de su participación en los ingresos corrientes de la Nación para subsidiar la adquisición de prótesis para la población en situación de discapacidad de escasos recursos, dentro de las atenciones del Plan Obligatorio de Salud [18].

Igualmente, el Ministerio de Trabajo y de Seguridad Social estableció, por medio del Decreto 1295, que todo trabajador que sufriera un accidente de trabajo o una enfermedad profesional tendría derecho a prestaciones asistenciales como prótesis y órtesis y rehabilitaciones física y profesional [19]. En el año 2018, se incluyen las demás instituciones, con la actualización del Plan de Beneficios en Salud, en donde se establecen las coberturas de los servicios y tecnologías en salud que deben ser garantizados por las Entidades Promotoras de Salud (EPS) o las entidades que hagan sus veces, a los afiliados al Sistema General de Seguridad Social en Salud (SGSSS), financiando prótesis ortopédicas externas (exoprótesis), para miembros superiores, incluyendo su adaptación, así como el recambio por razones de desgaste normal, crecimiento o modificaciones morfológicas del paciente [20].

Las prótesis de miembro superior pueden dividirse en 3 tipos, dependiendo de la función que cumplen en el usuario: cosméticas, mecánicas y electrónicas [7], [10], [11], [14]. Las prótesis cosméticas o pasivas tienen la ventaja de tener una apariencia muy similar a la mano natural, tienen bajo peso y requieren poco mantenimiento, sin embargo, no son funcionales. Las prótesis mecánicas aprovechan el movimiento de alguna parte del cuerpo o del miembro residual para generar el movimiento de la prótesis, son duraderas y funcionales; no obstante, en amputaciones transhumerales o transradiales pueden causar lesiones en el hombro debido a su uso prolongado. Las prótesis electrónicas se activan mediante señales musculares del miembro residual, permiten actividades de mayor precisión, tienen apariencia robótica; pero, en la mayoría de los casos tienen limitaciones en el peso que pueden cargar. También existen prótesis híbridas. las cuales son combinaciones de las prótesis anteriormente mencionadas (e.g. mecánicas + estéticas, mecánicas + robóticas, etc.) [10]. A pesar de que son muchas las funciones que pueden recuperarse con estas prótesis, estas presentan altas tasas de rechazo primario, definido como no uso de prótesis o de rechazo secundario, que se define como falta de continuidad en la utilización de la prótesis. En el estudio de Ostlie et al., se encontró que las principales razones para la no utilización primaria son la falta de necesidad percibida y las discrepancias entre esta necesidad y las prótesis disponibles [21]. En la literatura se ha reportado falta de adherencia a las prótesis de miembro superior por parte de los amputados tan alta como del 50% para ganchos mecánicos, 53% para manos pasivas y 39% para manos mioeléctricas [22], este rechazo se ha atribuido, principalmente, al elevado peso, la falta de confort y a la funcionalidad limitada de la prótesis (relacionadas con los mecanismos de acción de la misma), el alto costo, la limitación del uso de cierto tipo de ropa, irritaciones en la piel, aumento de temperatura en las zonas de contacto, la baja duración y la resistencia mecánica de la prótesis, la dificultad en el control, su apariencia estética, la falta de retroalimentación sensorial, la falta de educación, la falta de entrenamiento y la poca destreza [22]-[25]. Aunque son muchas las quejas que los usuarios tienen de su prótesis, se ha encontrado que los factores principales que deben modificarse para mejorar la aceptación de la prótesis son el funcionamiento, el confort y el control [21], [26].

El empleo de una prótesis con un resultado funcional favorable ha demostrado que lleva a una mayor cantidad de horas de uso al día, lo que permite una mejor interacción con el medio físico y el ambiente psicosocial que rodea a la persona con este tipo de amputación [23]. Además, el abordaje de las necesidades, prioridades o preferencias de los pacientes en cuanto al diseño de las prótesis es una forma de detectar aquellos factores que pueden influir en el rechazo de estos dispositivos y de superponerse a ellos. Un estudio de Biddiss *et al.* [27] encontró que la participación de los pacientes en la selección de la prótesis y la necesidad percibida de una prótesis son factores clave relacionados con la aceptación de este tipo de dispositivos. Es por ello que, para aumentar las tasas de aceptación de prótesis, las recomendaciones clínicas deben centrarse en estrategias de adaptación oportunas y en el desarrollo de prótesis y atención médica óptimas y centradas en el paciente con amputación de extremidades [28]. Los esfuerzos deben dirigirse a optimizar la comunicación entre los pacientes, los protesistas, los diseñadores y los ingenieros para mejorar la calidad de la atención brindada al creciente número de personas con pérdida de extremidades [29].

Es importante resaltar que en países desarrollados, las terapias nuevas deben ser evaluadas en términos de su eficacia y efectividad para poder ser aceptadas en las regulaciones de los sistemas de salud y recomendadas para el reintegro del dinero por parte de aseguradoras de salud [30], ya que estudios, como los de usabilidad, entregan medidas altamente confiables y válidas [24]. A pesar de su importancia, son pocos los estudios que reportan resultados del uso de prótesis de miembro superior con amputados que además tengan validez externa, garanticen la objetividad de los resultados y tengan significancia estadística [30]; al igual que reportes de uso en el corto y el largo plazo, especificaciones mecánicas como la fuerza de agarre, aceptación de uso, reproducibilidad, funcionalidad y durabilidad [31], [32]. Así mismo, los estudios sobre prótesis fabricadas con impresión 3D, que es la tecnología usada por Prótesis Avanzadas S.A.S., solo se enfocan en su diseño, tanto mecánico como electrónico, y no en la evaluación de su funcionamiento [25], [31]–[46].

En los últimos años, el auge de la tecnología de impresión 3D ha posibilitado el diseño y la fabricación de dispositivos médicos, incluyendo prótesis de miembro superior. Su uso permite tener la flexibilidad necesaria para crear estrategias de ajuste de prótesis centradas en el paciente, lo cual aumenta el índice de aceptación de la prótesis y, por lo tanto, facilita un ajuste exitoso [21], [28], [47]. Esto se debe a que la impresión 3D permite la personalización bajo demanda, la fabricación en sitio, y la generación de bajos costos [48]. Actualmente, el costo de una prótesis mioeléctrica está por encima de las 30.000 libras esterlinas según lo reportado por Sime en 2019 [49], y entre 25.000 y 75.000 dólares según datos reportados por Kate *et al.* en 2016 [31]; sin embargo, gracias al uso de tecnologías como la impresión 3D, se abren otras opciones en el mercado como la que ofrece Prótesis Avanzadas S.A.S. con un costo de apróximadamente \$13.000.000.

En un estudio desarrollado por Duong *et al.* se compararon las capacidades funcionales y la eficiencia de una mano mioeléctrica impresa en 3D (*i.e. Limbitless*) y una disponible comercialmente (*i.e. i-limb*). Se encontró que la mano comercial es más eficiente que la impresa en 3D, pero que existe potencial para que las prótesis impresas en 3D se conviertan

en una opción viable [25]. En el estudio de Lee *et al.* se realizó una comparación similar y se mostraron como ventajas de la impresión 3D la reducción de los costos y tiempo de producción, y la reducción del peso de la prótesis [43].

Todo lo anterior muestra la evidente necesidad que tiene el país de crear productos que puedan ayudar a esta población a recuperar parte de su autonomía y que sean desarrollados pensando en sus necesidades y sus capacidades económicas. El objetivo de este proyecto es entonces rediseñar, implementar y evaluar la efectividad de una prótesis mioeléctrica transradial de buena calidad, enfocadas en la población amputada colombiana y que mejoren los índices de aceptación [21], [28], desarrollando estrategias que suplan el vacío de información rigurosa sobre aceptación y buen funcionamiento de las prótesis impresas en 3D a través de estudios de efectividad [23], [30]. De esta manera, no solo se benefician los usuarios, sino que se comienza a potenciar al país como un referente en tecnología e innovación, solucionando problemas en los que es uno de los mayores afectados.

#### **ESTADO DEL ARTE**

Esta revisión se enfoca en las prótesis mioeléctricas transradiales con las que se dispone actualmente en el mercado y las investigaciones científicas sobre temas relacionados con ellas.

## Opciones comerciales de prótesis mioeléctricas

Existen varias empresas en el mundo que se dedican a fabricar prótesis mioeléctricas transradiales. A continuación, se presentan los principales referentes comerciales.

## Ottobock

Empresa alemana que por más de un siglo se ha dedicado al diseño y fabricación de órtesis y prótesis para personas con discapacidad. Su objetivo es ayudar a estas personas a mantener o recuperar la libertad en sus movimientos a través de desarrollos tecnológicos innovadores y servicios personalizados [50].

En prótesis de miembro superior, la empresa cuenta con cuatro opciones en el mercado: la mano *Michelangelo*, la mano *Myofacil*, la opción para niños *Electrohand* y la mano *be-bionic*.

## Michelangelo

La mano Michelangelo recupera muchas de las funciones de la mano natural, que además cuenta con un diseño natural que se integra de forma armónica con el cuerpo del ser humano. La mano posee 7 tipos de agarre y una muñeca *AxonWrist* que permite los movimientos de flexión/extensión y rotación interna y externa. Los dedos están fabricados combinando materiales duros y blandos para imitar la mano natural. Esta mano está cubierta con un guante protésico que viene en 6 colores diferentes [51].



Figura 1. Prótesis Michelangelo de la empresa Ottobock [51].

# MyoFacil

La prótesis *MyoFacil* es ideal para comenzar una adaptación con tecnología mioeléctrica. Está diseñada para realizar actividades al interior del hogar o en la oficina. Puede usarse en modo electrónico o de forma pasiva, dependiendo de lo que el usuario requiera [52].



Figura 2. Prótesis MyoFacil de la empresa Ottobock [52].

## Electro hand

Es una mano mioeléctrica diseñada especialmente para niños. Su tamaño es más pequeño y su peso más liviano que las opciones para adultos. El diseño de los dedos pulgar e índice permite agarrar utensilios para comer y escribir de una manera natural. Las manos vienen cubiertas con guantes de colores naturales que asemejan la piel u otros fuertes como rosado, rojo, azul y negro [53].



**Figura 3.** Prótesis *Electrohand* de la empresa *Ottobock* (izquierda). Mecanismo de agarre de la prótesis *Electrohand* (derecha) [53].



Figura 4. Cubiertas de colores para la prótesis Electrohand [53].

## Be-bionic

Es una mano artificial que ha sido diseñada para apoyar al usuario en el desarrollo de muchas de las actividades de la vida diaria: desde comer y cargar paquetes hasta abrir puertas y escribir en el computador. Está fabricada con materiales avanzados y duraderos que permiten cargar hasta 45 kg. Cuenta con motores individuales en cada dedo, lo que posibilita tener 14 tipos diferentes de agarre. La velocidad de cierre de la mano es proporcional a la contracción muscular, lo que da precisión para actividades delicadas y a la vez permite desarrollar actividades que requieren más fuerza. Está disponible en 3 tallas diferentes y con 4 opciones de muñeca, para acomodarse a los requisitos particulares del usuario. La mano posee una función llamada "Auto grip", que detecta de forma automática cuando un objeto se está deslizando y ajusta la mano para hacer el agarre más seguro [54].



Figura 5. Prótesis Be-bionic de la empresa Ottobock [54].

# **Touch bionics**

Touch Bionics es una empresa proveedora de tecnología protésica que hace parte de Össur, líder en dispositivos protésicos y ortésicos [55]. Cuenta con dos opciones de prótesis para miembro superior: *i-limb ultray i-limb quantum*. Con cualquiera de estas prótesis, los usuarios tienen derecho al programa *Touch Care Program*, que incluye garantía, cubrimiento por daños accidentales, app para el control de la prótesis, guante para la prótesis, chequeo médico, mano de cortesía mientras la propia está siendo arreglada, entrenamiento de la prótesis por medio de la app.

#### i-limb ultra

Esta prótesis se ve y se mueve como una mano natural. Su sistema electrónico permite que las articulaciones de cada dedo se doblen para adaptarse a la forma del objeto que está

siendo agarrado; también, permite incrementar la fuerza del agarre en situaciones donde se requiera, tales como amarrarse los cordones o abrir un tarro de comida. Posee 14 tipos de agarres que pueden ser programados mediante una aplicación móvil y un modo "auto-grasp" para prevenir que los objetos se deslicen. Después de un periodo de inactividad, la mano se mueve automáticamente a una posición natural. La mano está disponible en 3 tallas (S-M-L) y puede cubrirse con guantes transparentes o negros (*i-limb skin active*) o que tengan apariencia humana (*i-limb skin natural*) [56].



Figura 6. Prótesis i-limb ultra de la empresa Touch Bionics [56].

## i-limb quantum

i-limb quantum tiene articulación independiente en cada dedo y permite 36 tipos diferentes de agarres que pueden pre-programarse y controlarse por 4 medios: gesto, app, contracción muscular y proximidad. Posee el modo "vari-grip" por el que puede modificarse la fuerza de agarre y el "auto-grasp" que previene el deslizamiento de los objetos. La mano está disponible en 3 tallas (S-M-L) y puede cubrirse con guantes transparentes o negros (i-limb skin active) o que tengan apariencia humana (i-limb skin natural) [57].



Figura 7. Prótesis i-limb quantum de la empresa Touch Bionics [57].

# **Mobius bionics**

Mobius bionis es una empresa productora de dispositivos médicos, los cuales se basan en el desarrollo de productos tecnológicos con alto componente de investigación. Para las personas amputadas de miembro superior desarrollaron el brazo *LUKE*, que traduce *Life Under Kinetic Evolution* [58].

## Brazo LUKE

Es una prótesis de brazo modular que puede ser configurada para diferentes tipos de amputación: transradial, transhumeral y desarticulación de hombro. Posee un sistema de control flexible que contiene entradas de varios dispositivos tales como sensores mioeléctricos e IMUs. Posee varios tipos de agarre que pueden pre-programarse según la actividad que se quiera desarrollar y la velocidad de cierre en cada uno de estos puede ser ajustado por el usuario. La muñeca combina movimientos de flexo-extensión y desviación ulnar/radial, que permiten agarrar objetos por encima de la cabeza o debajo de la cintura. Puede usarse en el exterior bajo condiciones de polvo y lluvia suave [58].



Figura 8. Prótesis LUKE de la empresa Mobius [58].

#### Exiii

Exiii es una compañía japonesa que desarrolló la prótesis handiii COYOTE, la cual fue pensada como una solución mioeléctrica funcional de bajo costo, que terminó costando menos de US\$ 300 [59].

# Handiii

La prótesis *Handiii* fue desarrollada teniendo como base 3 principios: 1. Que el procesamiento del sensor y los algoritmos de control se pudieran realizar en un smartphone regular, 2. Reducir el número de motores a 1 por dedo y no a uno por articulación y 3. Usar la impresión 3D para reducir los costos de manufactura, para permitir facilidad en la reparación y en la personalización [59].

El sensor de EMG usado en esta prótesis envía información de forma inalámbrica al Smartphone y éste interpreta esta señal para controlar el brazo. El tipo de agarre se escoge mediante un botón ubicado en el codo. Los aspectos más diferenciadores de este producto son su precio y su diseño estético [59].



Figura 9. Prótesis Handiii de la empresa Exiii [59].

#### **Pro-bionics**

*Probionis* es una Pyme nacida en México en el año 2006 cuyo campo de acción son las prótesis mioeléctricas de miembro superior y que cuenta con 5 patentes en Estados Unidos, Comunidad Europea y Brasil [60].

La prótesis consiste en un gancho electrónico modular que puede ser adaptada para amputaciones transradiales, desarticulaciones de codo, transhumerales y desarticulaciones de hombro para realizar tanto actividades que requieran cargar peso como otras que requieran movimientos finos. Tiene la opción de ser cubierta con un guante cosmético que asemeja la apariencia humana de la mano [60].





Figura 10. Prótesis de miembro superior de la empresa Probionics [60].

# Vincent Systems

Vincent Systems es una empresa dedicada a avances en tecnología médica, en especial a la producción de prótesis con alto contenido de innovación. Para amputaciones transradiales, esta empresa ofrece la opción *VINCENTevolution* [61].

# VINCENTevolution

Esta prótesis combina funcionalidad y calidad con bajo peso. Está fabricada con acero inoxidable y con una aleación de alta resistencia de magnesio-aluminio. Posee 6 motores que permiten el movimiento independiente de cada dedo y la posibilidad de escoger entre 14 tipos de agarres diferentes. La sujeción de objetos es fácil, gracias a la precisión de los dedos pulgar e índice y que los pulpejos tienen superficies planas. Cuenta con una app para que el usuario pueda entrenarse en el control del sistema. El usuario puede escoger entre diferentes tallas y puede decidir usarla con o sin guante cosmético [61].



Figura 11. Prótesis VINCENTevolution de la empresa Vincent Systems [61].

#### Prótesis mioeléctricas en literatura científica

La mayoría de los casos reportados sobre prótesis de miembro superior en revistas científicas mencionan diseños elaborados en impresión 3D en los que sólamente se comprueba la funcionalidad del diseño; mientras que las prótesis que se encuentran disponibles en el mercado carecen de estudios científicos que tengan validez externa, garanticen la objetividad de los resultados, tengan significancia estadística [30] y reporten resultados de uso tanto en el corto como en el largo plazo [31], [32].

Los *reviews* más recientes sobre prótesis de miembro superior en impresión 3D concluyen sobre el alto nivel de reducción de costos en la personalización de las prótesis de miembro superior impresas en 3D, pero señalan los desafíos que deben ser enfrentados sistemáticamente; como la durabilidad, una fuerza de sujeción suficiente, la reproducibilidad, y un atractivo general para la mayoría de los usuarios. Vujaklija *et al.* consideran que la introducción de nuevos materiales para impresión pueden ayudar a superar algunos de estos problemas, pero se debe tener presente el riesgo adicional que se tiene con estos nuevos materiales, ya que pueden aumentar los costos y disminuir la disponibilidad de las prótesis [32].

Así mismo, en un *review* de 2016 [31] donde se toma en consideración la información cuantitativa reportada, identifican que:

- Más de la mitad de las prótesis transradiales reportadas tienen alimentación externa, estas en su mayoría son controladas a través de electromiografía, con algunas pocas controladas por electroencefalografía y voz.
- Los costos son de entre 5 dólares y 500 dólares, pero ninguna de las prótesis puede ser comprada a un proveedor; se pueden encontrar algunos proveedores que ofrecen prótesis entre 1.000 dólares y 3.000 dólares, como You Bionic (200 dólares según precios actuales) y Open Bionics (entre 150 y 520 libras esterlinas según precios actuales). Más de la mitad de los diseños reportados en la literatura se encuentran como código abierto en distintas plataformas.
- Los pesos reportados incluyen una prótesis de 71 g desarrollada por M. Groenewegen y la *Roboarm* desarrollada por *Unlimited Tomorrow* que pesa 2.000 g (aunque es un brazo completo, no incluye el peso de los elementos electrónicos); el resto pesan entre 132 g y 960 g, con la mayoría en un rango entre 240 g y 450 g.

- No hay evidencia de su aceptación, funcionalidad o durabilidad. Y, aunque la impresión 3D no siempre es más económica, muestra posibilidades prometedoras para la personalización (e.g. socket personalizado, color, tamaño) sin ser necesario el ajuste de los equipos de producción.
- La mayoría fueron impresas en 3D usando Modelado por Deposición Fundida (FDM), seguidas por las impresas por (Sinterizado Láser Selectivo) SLS, y solo una prótesis reportada usando Estereolitografía (SLA) y una usando PolyJet.

Con respecto a los estudios más recientes sobre el uso de impresión 3D para la creación de prótesis de miembro inferior se tienen desde metodologías de diseño que se soportan en la impresión 3D para la fabricación de las prótesis, y prótesis fabricadas a través de esta tecnología en las que solo se evalúa su funcionalidad. Por ejemplo, Cabibihan *et al.* [45] presentó una metodología en la que se recreó la forma y tamaño del brazo amputado con una alta exactitud a través de impresión 3D y modelado de silicona. El proceso de fabricación de la prótesis puede observarse en la Figura 12 y el del socket en la Figura 13.



**Figura 12.** Proceso de diseño y fabricación del brazo protésico que implica el uso de imágenes tomográficas del brazo sano, el cual fue usado como base para la creación del molde con el que se fabricó la prótesis en silicona [45].



**Figura 13.** Proceso de diseño y fabricación del socket, que incluye la impresión 3D del miembro residual para ser usado como molde positivo en la fabricación del socket a través de los métodos tradicionales [45].

Ejemplos de diseños desarrollados en los últimos años se encuentran en los trabajos de Ariyanto *et al.* [41], Fajardo *et al.* [42], y Curline-Wandl *et al* [44]. El diseño de Ariyanto *et al.* [41] emplea un actuador lineal combinado con mecanismos de tendones-resortes, cinco modos de agarre para permitir actividades de la vida diaria, y controla los movimientos de flexión y extensión de la mano. La prótesis *AstoHand* desarrollada puede observarse en la Figura 14.



**Figura 14.** *AstoHand* V3.0 implementada en el estudio con un participante con amputación transradial [41].

Así mismo, se tiene el diseño de la mano Galileo, desarrollada por Fajardo et al. [42], el cual es un diseño simple pero funcional, realizado a través de impresión 3D con el fin de reducir costos y ahorrar tiempo en el proceso de manufactura. Este es también un diseño modular, paramétrico y autocontenido que busca ajustarse a un amplio rango de personas con amputación transradial en diferentes niveles, su control por medio de electromiografía de superficie permite al usuario activar conscientemente el mecanismo actuador de la prótesis, y una interfaz gráfica da la posibilidad de seleccionar entre un conjunto de gestos predefinidos. En la Figura 15 se puede observar el diseño de la mano Galileo.



Figura 15. Mano Galileo, versión biónica impresa en 3D, de 15 grados de libertad y subactuada [42].

Curline-Wandl *et al.* [44] presenta una investigación piloto sobre el uso de impresión 3D y un microprocesador Arduino de bajo costo como una alternativa económica a los dispositivos de alto costo, que además se enfoca en desarrollar una prótesis de bajo peso, fácil de controlar, y que tenga una morfología similar a la mano humana. Este diseño se puede observar en la Figura 16.



Figura 16. Modelo de impresión 3D de la Talonhand 2.7 [44].

También se han desarrollado trabajos a niveles de pregrado con el fin de diseñar prótesis mioeléctricas. En este caso, una mano impresa en 3D fue diseñada con una funcionalidad sofisticada; un socket ajustable y cómodo; de bajo peso, pero resistente; disponible a un precio razonable [46].



Figura 17. Prototipo desarrollado como trabajo para obtener el título de pregrado [46].

Finalmente, existen enfoques más innovadores como el de la *SoftHand Pro* (SHP). La SHP es una mano protésica funcional y robusta que minimiza costo y peso usando un diseño subactuado con un solo motor. Luego de pruebas, se estableció que esta prótesis es fácil de usar, al mostrar grandes mejoras luego del entrenamiento; además de no encontrarse diferencia en la mayoría de medidas clínicas de desempeño al compararla con dispositivos comerciales; excepto en abotonarse una camisa y usar el celular, donde mostró mejores resultados; y en la manipulación de objetos pequeños donde mostró peores resultados [33]. En la Figura 18 se puede ver el diseño de la SHP.



**Figura 18.** A: La SoftHand Pro (SHP) con una interfaz en la muñeca. B: La SHP agarrando un tubo cuadrado grande, con ventaja debido a su diseño de articulaciones flexibles. SHP demostrando capacidades de giro (C), doblez (D) y desarticulación (E, F) [33].

Además de los nuevos diseños de prótesis transradiales, varios investigadores han trabajado en mejorar el análisis de las señales mioeléctricas, ya que aunque las prótesis controladas vía electromiografía superficial representan la solución más avanzada y no invasiva para restaurar el funcionamiento de la mano de amputados de miembro superior, aún presentan dificultades en su control [36]. Por ejemplo, existen varias técnicas de electromiografía que permiten clasificar los movimientos de manos. Waris *et al.* [38] comparó entre las técnicas de: análisis discriminante lineal, red neuronal artificial, máquinas de vectores de soporte, k vecinos más próximos y árbol de decisión; encontrando que la red neuronal artificial presenta la clasificación de exactitud más alta, seguida por el análisis discriminante lineal.

Así mismo, Iqbal *et al.* [34] mejoró el desempeño en los movimientos de flexión y agarre de prótesis mioeléctricas, entre un 7% y un 9%, al usar técnicas no lineales para analizar las señales electromiográficas (las cuales son señales no lineales y no estacionarias). Con las técnicas no lineales logró que el sistema se adaptara mejor a las variaciones en los niveles de contracción de los músculos, lo que impactó positivamente el reconocimiento de patrones basados en el control mioeléctrico. Mientras que Schmalfuss *et al.* [37] desarrolló un enfoque híbrido, con un segundo grado de libertad controlado por la actividad mioeléctrica de los músculos auriculares posteriores; además del control convencional en el antebrazo. Este enfoque mostró que los sujetos controlaban la prótesis más rápidamente y más exactamente, y la robustez del sistema no se vio comprometida por las diferentes posiciones del brazo. Lo anterior permite tener un control más sofisticado, que se adapta las condiciones de la vida real, a diferencia de los esquemas de control tradicionales.

Como trabajos alternos, se ha explorado el uso de una banda de brazo de bajo costo para reconocimiento de gestos llamada Myo, la cual es capaz de identificar cinco gestos de mano, mostrando capacidad para ser usada como sistema de control mioeléctrico. Este estudio, realizado por Cognolato et al. [36], evaluó el desempeño de la Myo en amputados de mano, y los cuatro gestos de mano analizados mostraron resultados entre el 50% y 97% de precisión También existen estudios basados en la retroalimentación intraneural sensorial. la cual mejora el control sensomotor que tiene el amputado transradial de su prótesis mioeléctrica [39]. Aunque varios grupos de investigación han logrado tener retroalimentación táctil en amputados de miembro superior usando electrodos implantados, estimulación de nervios superficiales o substitución sensorial; el estudio de D'Anna et al. [40] demostró que se podía obtener información táctil a través de la simulación neural somatotópica e información de propiocepción a través de substitución sensorial, de manera simultánea y eficiente. Otro ejemplo de desarrollos recientes es el estudio de Clemente et al. [39], donde se llevaron a cabo distintas pruebas con una paciente y se midió su habilidad para regular finamente la fuerza de agarre aplicada; la paciente fue capaz de generalizar y transferir las habilidades de manipulación a otra tarea desconocida y mejorar su coordinación motora.

# CARÁCTER NOVEDOSO DE LA TECNOLOGÍA O PRODUCTO

A través de este proyecto se buscar desarrollar mejoras sustanciales en la prótesis mioeléctrica actual con la que cuenta la empresa Prótesis Avanzadas. Actualmente, el producto ofrecido por la empresa es el único de estas características producido a nivel nacional (manejo de la prótesis a través de sensores mioeléctricos), que además tiene un precio muy competitivo cuando es comparado con los precios de las prótesis importadas, y tiene una calidad superior si se compara con las prótesis de código abierto que se encuentran disponibles y que son usadas por fundaciones sin ánimo de lucro para su donación.

El objetivo principal de este proyecto es desarrollar una prótesis con un menor nivel de rechazo, ya que como se mencionó anteriormente, las prótesis de miembro superior presentan bajos índices de adherencia. Se espera lograr esto realizando cambios que ya han sido detectados como necesidades de los usuarios de las prótesis, como el uso de tecnologías de impresión 3D de alta gama, que permitan ensambles más eficientes y materiales más resistentes, que además lleven a un diseño que permita actividades de alto desempeño por los usuarios. Esta tecnología de impresión 3D también permitirá la fabricación de sockets con un ajuste cómodo, que se adaptará a los cambios de volumen del miembro residual. Finalmente, la inclusión en la etapa de diseño de los usuarios y diferentes personas involucradas en el proceso de adaptación de una prótesis mioeléctrica ha probado ser una estrategia efectiva para el aumento de la adherencia; por lo que se espera que al incluirlos realicen otras mejoras que aumenten la adherencia.

#### **OBJETIVOS**

# **Objetivo General**

Construir y validar pre-comercialmente una prótesis mioeléctrica para mejorar el funcionamiento de personas con amputación transradial.

## **Objetivos Específicos**

- 1. Establecer los nuevos requerimientos técnicos de las prótesis transradiales mioeléctricas y seleccionar el concepto de diseño que mejor cumpla con estos requerimientos.
- 2. Definir el diseño de detalle de las nuevas prótesis transradiales mioeléctricas, garantizando el cumplimiento de los criterios técnicos y económicos de éstas.
- Evaluar la efectividad de las nuevas prótesis transradiales mioeléctricas a partir de prototipos, en comparación con el no uso, para mejorar el funcionamiento de personas con amputación transradial.
- 4. Realizar el análisis financiero de la nueva prótesis mioeléctrica transradial, incluyendo aspectos económicos y comerciales.

# METODOLOGÍA Y PLAN DE TRABAJO DEL PROCESO DE VALIDACIÓN PRE-COMERCIAL

La metodología para el resideño de la prótesis mioeléctrica transradial buscará adicionar valor al diseño actual, al aumentar el valor percibido por el comprador proporcionando atributos adicionales a los actuales. La metodología se dividirá en cinco fases principales que van desde la clarificación de los objetivos que se esperan satisfacer con el diseño, hasta la creación y evaluación de un prototipo funcional que haya sido mejorado luego de la realización de pruebas de desempeño, y realizando una evaluación de efectividad, además de una fase paralela a todas que incluye el análisis financiero. El detalle de cada una de las fases se encuentra a continuación.

# Diseño conceptual

Durante esta fase se buscará definir el concepto sobre el que se va a desarrollar el rediseño de la prótesis transradial basado en el Método de Diseño de Cross [62]. Inicialmente, se deberá hacer un planteamiento completo y claro de los objetivos que debe satisfacer la prótesis a través de la *clarificación de objetivos*. Luego, se continuará con el *establecimiento de funciones*. A partir de la identificación del nivel de generalidad o detalle en el que se va a trabajar, se definirán las funciones y los límites del problema a solucionar, estableciendo las funciones específicas que debe satisfacer la prótesis, independientemente de los componentes físicos que pudieran utilizarse.

Posteriormente, se procederá con la *fijación de requerimientos*, en donde se definirá la especificación del rendimiento de la prótesis, lo cual permitirá evaluar que las soluciones propuestas se encuentren dentro de los límites aceptables. Además, se elaborará la *determinación de características*, donde se compararán los atributos deseables del nuevo producto - desde el punto de vista del cliente - con los requerimientos de ingeniería definidos previamente. Esta comparación se realizará a través del despliegue de la función de calidad lo cual implica entrevistas o encuestas a posibles usuarios y expertos en el tema, sesiones de grupo, búsqueda del estado del arte, entre otros.

Finalmente, se llevará a cabo la *generación de alternativas* y su *evaluación*. La *generación de alternativas* se basa en el método del diagrama morfológico, el cual presenta la gama completa de elementos, componentes o soluciones secundarias que pueden combinarse para formar distintas soluciones, a partir de los cuales se definirán los diseños alternativos. Durante

la evaluación de alternativas se valorarán los diferentes diseños alternativos de acuerdo a los requerimientos y objetivos definidos previamente.

Para estas actividades, se contará con un grupo de participantes con amputación transradial que acepten ingresar al estudio. En la sesión se evaluarán, de manera cualitativa, las prioridades y preferencias de los pacientes con respecto al uso de prótesis y a las necesidades que éstas deberían cubrir. Se indagará por aspectos como la usabilidad, el confort, la adaptación, la fuerza, la movilidad, el desempeño en las actividades de la vida diaria y la calidad de vida [24].

Adicionalmente, se buscará con la participación de profesionales involucrados en la rehabilitación de los pacientes con amputación de miembro superior, a quienes también se entrevistará para definir los objetivos y los aspectos clínicos a tener en cuenta en el diseño de la prótesis. Así mismo, ambas entidades (Prótesis Avanzadas y la Universidad de Antioquia) conservarán los entregables de esta fase del diseño.

#### Diseño de materialización

Esta fase del diseño sigue la metodología establecida para el Diseño en Ingeniería por Pahl y Beitz [63], y en ella se desarrolla el diseño de la prótesis mioeléctrica transradial a partir del concepto definido en la fase anterior y teniendo en cuenta los criterios técnicos y económicos del mismo. Además, debe llevar al diseño definitivo de las prótesis, luego de verificar que el funcionamiento, durabilidad, producción, ensamble, operación y costos del diseño cumplen con las especificaciones.

Es importante tener en cuenta que debido a la complejidad del diseño de materialización (*i.e.* algunas actividades se deberán repetir cuando se tenga mayor información, los cambios realizados en un área del diseño pueden afectar otras, varias acciones deben llevarse a cabo simultáneamente), problemas particulares que se encuentren pueden generar desviaciones sobre lo planeado. Por lo tanto, se recomienda desarrollar esta fase partiendo de lo más general a lo más específico y definiendo puntos de verificación para realizar correcciones. Entre las actividades a realizar se encuentran:

- Establecer cuáles funciones tienen impacto directo en la determinación del tamaño de las prótesis.
- Determinar cuáles funciones deben satisfacerse en conjunto.
- Definir los bocetos detallados de acuerdo a normas, estándares, cálculos detallados o resultados experimentales.
- Evaluar los bocetos con respecto a los criterios técnicos y económicos.

Ambas entidades conservarán los entregables de esta fase del diseño.

## Diseño de detalle

En esta fase del diseño se espera obtener los documentos necesarios para la producción de las prótesis mioeléctricas. En nuestro caso específico, debido a que el sistema de producción de Prótesis Avanzadas se basa en la impresión 3D, los documentos principales serán los archivos CAD de los componentes diseñados, la lista de partes que incluya tanto los elementos comerciales como los componentes impresos, el plano de ensamble y el manual de uso de la prótesis. Ambas entidades conservarán los entregables de esta fase del diseño.

# Evaluación pre-comercial

Como fase final del diseño se procederá a la fabricación de un prototipo y la realización de pruebas de desempeño del mismo. Así mismo, se realizarán pruebas de producción en las que se identifiquen problemas con la creación de las prótesis. Finalmente, con los resultados de las pruebas, se procederá a desarrollar las mejoras del diseño, actualizando los documentos necesarios para la producción de las prótesis y obteniendo un prototipo del diseño mejorado. Una vez definido el diseño se realizará un estudio de efectividad con pacientes con amputación transradial.

#### Diseño del estudio de efectividad

Se realizará un ensayo clínico con diseño cruzado aleatorizado para definir el momento de la intervención en doce participantes. Este tipo de diseño reduce la influencia de las variables de confusión porque los sujetos pueden actuar como su propio control en el ensayo [64], [65] y son ideales para evaluar intervenciones en condiciones crónicas y estables, como es el caso de las amputaciones de extremidades [24].

En la Figura 19 se muestra el diseño propuesto. Se compararán entonces la intervención, es decir el uso de la prótesis mioeléctrica versus el no uso de la prótesis. Se asume que no hay efecto de "arrastre" pues se espera que la intervención (prótesis) tenga el efecto deseado mientras se utiliza y que no tenga un efecto residual en el funcionamiento al retirarla, por lo tanto, no se requiere periodo de lavado entre las intervenciones.



Figura 19. Esquema ejemplo del diseño del estudio.

#### Población

La población de referencia y de estudio serán pacientes adultos con amputación transradial unilateral de cualquier causa.

# Criterios de inclusión

- Que vivan en Medellín o el área metropolitana y puedan desplazarse al lugar de evaluación
- Pacientes que sean capaces de comprender y seguir órdenes.

#### Criterios de exclusión

- Pacientes con amputación bilateral de miembros superiores.
- Pacientes con lesiones en piel o tejidos blandos que contraindiquen el uso de prótesis.

## Selección y tamaño de la muestra

El muestreo se realizará por conveniencia y los pacientes se seleccionarán de la consulta de fisiatría, cirugía plástica u ortopedia de las instituciones participantes. El número de pacientes se seleccionó teniendo en cuenta los costos del diseño, los costos y tiempo requerido para la elaboración de las prótesis, el tiempo requerido para las pruebas de efectividad y los recursos disponibles para el proyecto.

# Intervención y control

Cada prótesis será entregada por integrantes del equipo de diseño y una terapeuta física u ocupacional, quienes realizarán los ajustes necesarios para la adaptación y entrenarán en el uso de ésta durante dos sesiones de 3 horas cada una. En el grupo de intervención los pacientes usarán la prótesis durante un periodo de dos semanas y luego de este tiempo se citarán para la aplicación de las escalas de funcionamiento, satisfacción y calidad de vida. Los pacientes asignados al grupo control serán citados para la aplicación de las escalas de funcionamiento y calidad de vida. Los controles se realizarán sin el uso de la prótesis pues este es el escenario más común en los amputados de miembro superior y queremos demostrar que el uso de prótesis es superior al "no tratamiento".

No se requiere periodo de "lavado" (*washout*) entre los periodos ya que se espera que la intervención (prótesis) tenga el efecto deseado mientras se utiliza y que no tenga un efecto residual al retirarla. No será posible realizar cegamiento de los participantes o los investigadores debido al tipo de intervención y de medición de desenlaces.

## Desenlaces

Para este estudio, se seleccionaron desenlaces se evaluarán: el funcionamiento definido como desempeño en actividades cotidianas, tanto autorreportado como observado; la satisfacción con la prótesis y la calidad de vida relacionada con la salud (Tabla 1). Recientemente, el Grupo de trabajo sobre medidas de resultados protésicos de extremidades superiores (ULPOM) recomendó el uso de la Clasificación Internacional de Funcionamiento, Discapacidad y Salud (CIF) de la Organización Mundial de la Salud como marco ideal para seleccionar los instrumentos y desenlaces, y destacó la importancia de seleccionar las herramientas de evaluación que tuvieran en cuenta cada uno de los elementos importantes de la CIF, incluidas las estructuras y funciones corporales (rendimiento de la prótesis), la actividad (realizar tareas) y la participación (uso de la prótesis en situaciones de la vida real) [66].

**Tabla 1.** Desenlaces e instrumentos para medirlos.

| Desenlace | | Instrumento | Número de<br>mediciones | Fuente |
|---|---|---|---|---|
| Funcionamiento<br>(Desempeño<br>actividades) | en | Orthotics and Prosthetics<br>Users Survey - Upper<br>extremity Functional status<br>(OPUS – UEFS) | 2 en cada<br>paciente | Autorreporte de pacientes |
| Funcionamiento<br>(Desempeño<br>actividades) | en | Brief activity performance<br>measure for upper limb<br>amputees (BAM-ULA) | 2 en cada<br>paciente | Observado por investigador |

| Desenlace | Instrumento | nto Número de mediciones | |
|---|---|---|---|
| Satisfacción con la prótesis | Orthotics and Prosthetics<br>Users Survey - Satisfaction | 2 en cada<br>paciente (solo<br>durante el uso<br>de prótesis) | Autorreporte de pacientes |
| Calidad de vida<br>relacionada con la<br>salud | Orthotics and Prosthetics<br>Users Survey - Health Quality<br>of Life Index | 2 en cada<br>paciente | Autorreporte de pacientes |

# Variables

En el instrumento se incluirán características sociodemográficas de los participantes como edad, sexo, estado civil, nivel educativo, ocupación. Además, se registrarán datos clínicos como tiempo desde la amputación, dominancia, mano afectada. La Tabla 2 resume la información sobre la operacionalización de estas variables.

Tabla 2. Operacionalización de las variables.

| Nombre<br>de la<br>variable | Nombre completo y unidad de medida | Naturaleza | Nivel de<br>medición | Código |
|---|---|---|---|---|
| edad | Edad del paciente en años | Cuantitativa | Razón | Años |
| sexo | Sexo del paciente | Cualitativa | Nominal | 0 Femenino<br>1 Masculino |
| ecivil | Estado civil | Cualitativa | Nominal | 0 Soltero<br>1 Casado<br>2 Unión libre<br>3 Viudo<br>4 Separado |
| neduc | Nivel educativo | Cualitativa | Nominal | O Primaria incompleta Primaria completa Secundaria incompleta Bachiller Profesional Técnico Tecnólogo Posgrado |
| ocupac | Ocupación | Cualitativa | Nominal | Empleado Independiente Pensionado |
| tiempo | Tiempo desde la amputación en meses | Cuantitativa | Razón | Meses |
| dominan | Mano dominante | Cualitativa | Nominal | 0 Derecha<br>1 Izquierda |
| manoaf | Mano afectada | Cualitativa | Nominal | 0 Derecha<br>1 Izquierda |
| opusuefs | Funcionamiento medido con la escala OPUS UEFS | Cuantitativa | Intervalo | Puntaje |
| bamula | Funcionamiento medido con la escala BAM-ULA | Cuantitativa | Intervalo | Puntaje |
| opussatis | Satisfacción con la prótesis con la escapa OPUS Satisfaction | Cuantitativa | Intervalo | Puntaje |

| Nombre<br>de la<br>variable | Nombre completo y unidad de medida | Naturaleza | Nivel de<br>medición | Código |
|---|---|---|---|---|
| opusqol | Calidad de vida<br>relacionada con la salud<br>con la escala OPUS<br>Health Quality of Life<br>Index | Cuantitativa | Intervalo | Puntaje |

#### Instrumentos

Se medirán desenlaces con cinco instrumentos, los cuales se encuentran como archivos anexos:

Instrumento para la recolección de datos demográficos

Diseñado por los investigadores para este proyecto (Ver Anexo 1. F-01 Formulario recolección).

Orthotics and Prosthetics Users Survey - Upper Extremity Functional Status (OPUS – UEFS) La Escala funcional de extremidades superiores (UEFS) es una de las escalas de la Encuesta de usuarios de prótesis y ortesis (OPUS) [67], [68] que ha demostrado ser confiable [68], [69]. El OPUS UEFS es la única medida autoreportada del desempeño de la actividad desarrollada específicamente para adultos con amputación de extremidades superiores. Es un instrumento para reportar la dificultad o facilidad en la ejecución de 23 tareas de la vida diaria y autocuidado [70]. Las tareas se califican en una escala de 1 a 5 puntos (desde muy fácil hasta no puedo realizar la actividad), independientemente de cómo se realicen las actividades (con o sin una prótesis). Las puntuaciones van de 0 a 100, las más altas indican más dificultad en la realización de actividades. La mayoría de los cuestionarios reportados por los pacientes toman menos tiempo en comparación con las medidas de observación. En el estudio se pedirá al paciente que puntúe el cuestionario según la realización de actividades con y sin la prótesis, dependiendo del momento de intervención. Este instrumento no se encuentra traducido ni validado para el español, se utilizará una versión traducida por los investigadores para este proyecto (ver Anexo 2. F-02 OPUS Estado funcional).

# Brief activity performance measure for upper limb amputees (BAM-ULA)

Es una medida observacional del desempeño en actividades [70]. Las diez actividades incluidas en el instrumento son: meter la camisa en los pantalones; levantar una bolsa de 20 libras; abrir una botella de agua; sacar una billetera del bolsillo trasero del pantalón; devolver la billetera al bolsillo trasero del pantalón; tomar una jarra de agua de un galón del refrigerador y ponerla en el mesón; verter agua de una jarra de un galón en un vaso; cepillar o peinar el cabello; usar un tenedor y abrir una puerta con pomo. Cada ítem se califica desde cero cuando "no se puede completar" o uno para "se completó". Las puntuaciones de cada elemento se suman para obtener la puntuación general de finalización de la tarea. Las puntuaciones de resumen se calculan sólo cuando se califican los diez elementos. Las puntuaciones más altas en la finalización de las actividades indican un mejor rendimiento. Los análisis de las propiedades psicométricas en una muestra de personas con amputación de extremidades superiores mostraron que el BAM-ULA tiene una consistencia interna aceptable, una fiabilidad test-retest y muestra evidencia de validez de constructo y concurrente [70]. Este instrumento no se encuentra traducido ni validado para el español, se utilizará una versión traducida por los investigadores para este proyecto (ver Anexo 3. F-05 BAM ULA Función).

# Orthotics and Prosthetics Users Survey – Satisfaction

Esta otra escala del OPUS mide la satisfacción del paciente con el dispositivo y con los servicios [67]. Se evalúan ítems sobre las características del dispositivo como "el peso de mi prótesis (u ortesis) es manejable" y "mi prótesis (u ortesis) es duradera"; características del uso del dispositivo como " mi prótesis (u ortesis) es fácil de colocar" y "mi ropa está libre de desgaste por la prótesis (u ortesis)"; y complicaciones asociadas al uso del dispositivo "mi piel está libre de abrasiones e irritaciones" y "el uso de mi prótesis (o la ortesis) es libre dolor". Este instrumento no se encuentra traducido ni validado para el español, se utilizará una versión traducida por los investigadores para este proyecto (ver Anexo 4. F-03 OPUS Satisfacción).

# Orthotics and Prosthetics Users Survey - Health Quality of Life Index

El puntaje de calidad de vida en salud del OPUS consta de 23 elementos que evalúan la calidad de vida relacionada con la salud. Los ítems incluyen: "¿con qué frecuencia durante la semana pasada ha estado feliz?"; "¿en qué medida su condición física restringe su capacidad para hacer tareas? [69]. Los ítems se evalúan en una escala de calificación de 5 puntos. El puntaje total del instrumento se calcula sumando de los puntajes de los 23 ítems. Una puntuación más alta indica un mejor resultado. Las preguntas de los instrumentos del OPUS se centran en la participación del paciente en la toma de decisiones [71]. Este instrumento no se encuentra traducido ni validado para el español, se utilizará una versión traducida por los investigadores para este proyecto (ver Anexo 5. F-04 OPUS Calidad de vida).

## Plan de recolección de los datos

Para obtener los datos de los posibles participantes se contactará a pacientes que cumplan los criterios de inclusión, se enviarán invitaciones para ser parte del estudio, con un resumen del mismo y se planearán visitas luego de acordar citas con aquellos que hayan aceptado participar. En las visitas se confirmará el cumplimiento de los criterios de inclusión, se explicarán los objetivos y la metodología del proyecto y se obtendrá el consentimiento informado. Los datos se tomarán de fuentes primarias mediante la aplicación de instrumentos diligenciados por el participante e instrumentos de desempeño supervisados por uno de los investigadores. La asignación aleatoria se realizará mediante códigos generados por computador, en sobres cerrados y opacos. Se realizarán dos mediciones de los desenlaces, con y sin el uso de prótesis, separadas por un periodo de 2 semanas. Una persona será responsable de la recolección de los datos y deberá verificar la calidad de los registros y la presencia de datos faltantes antes de retirarse del lado del participante. El investigador principal revisará la calidad de los registros y la presencia de datos faltantes que requieran volver a contactar al participante de forma personal o telefónica.

Los datos obtenidos mediante la aplicación de los instrumentos serán digitalizados por uno de los investigadores y revisados por el investigador principal para controlar la calidad del dato. Se consignará todo en una base de datos en MS Access®.

#### Plan de análisis estadístico

Se determinarán las características de la muestra usando estadística descriptiva. Para las variables cualitativas (*i.e.* nivel educativo, sexo, estado civil, ocupación, dominancia, miembro afectado) se presentarán frecuencia absoluta y relativa expresada en porcentaje. Para los análisis estadísticos se usará un enfoque bayesiano, el cual está recomendado para las

pruebas clínicas con dispositivos médicos [72]. Se estimarán indicadores de funcionamiento de la prótesis en actividades de la vida diaria, usando métodos bayesianos de estimación para el grupo con uso de la prótesis y el mismo grupo sin uso de la prótesis. En este caso se obtendrán intervalos de credibilidad para las principales variables del instrumento *OPUS Upper extremity functional status* y se compararán los resultados en los dos grupos para determinar la diferencia, si es que existe. Se determinará la asociación entre los indicadores de funcionamiento con variables sociodemográficas a través de pruebas bayesianas.

Además. se describirán estadísticamente los indicadores de funcionamiento observados según las variables del instrumento BAM-ULA y se estimará la correlación entre el funcionamiento medido por el paciente amputado y el funcionamiento observado por el investigador. Y para el análisis de la información de calidad de vida, se obtendrán indicadores según la escala *OPUS Health Quality of Life Index* que permitirá establecer una caracterización de los pacientes y su calidad de vida percibida. Para esto se estimarán indicadores con puntajes globales a través de los intervalos de credibilidad bayesianos de la calidad de vida de estos pacientes. Finalmente, para evaluar la satisfacción de los pacientes con la prótesis, se estimará la satisfacción global según las variables del instrumento *OPUS Satisfaction* y se explorará la asociación de la satisfacción con variables sociodemográficas.

Todos los análisis estadísticos se llevarán a cabo usando métodos Bayesianos el software R.

#### Consideraciones éticas

Según la Resolución 8430 de 1993 [73] por la cual se establecen las normas científicas, técnicas y administrativas para la investigación en salud, se considera una investigación con bajo riesgo. Se buscará la aprobación de un Comité de Bioética de Investigación en Humanos.

La investigación en seres humanos debe estar regida por tres principios éticos básicos [74]. El principio de respeto por las personas, que se refiere a la autonomía en la participación de un estudio; se garantiza mediante el consentimiento informado y el respeto por la autonomía, aclarando que la participación es voluntaria y puede detenerse en cualquier momento del estudio. El principio de beneficencia se refiere al esfuerzo por promover el bienestar del sujeto de investigación buscando lograr el máximo beneficio con el mínimo de riesgo y daño. El principio de justicia se relaciona con la selección equitativa de los participantes y el acceso equitativo a los riesgos y beneficios.

El equipo investigador se compromete a cumplir las normas de buenas prácticas clínicas en investigación. Entregaremos información detallada a cada participante sobre el propósito e importancia del estudio y solicitaremos un consentimiento informado a cada uno. El equipo de investigación será responsable de la confidencialidad de los datos de los pacientes. Se codificará la información y se guardará bajo custodia. Al finalizar la investigación, el equipo se compromete a divulgar los resultados.

Cabe aclarar que las prótesis se clasifican como dispositivos médicos no invasivos y que la empresa Prótesis Avanzadas cuenta con experiencia en la producción de prótesis en impresión 3D para miembro superior.

#### Análisis financiero

Para poder analizar la viabilidad financiera de la nueva prótesis mioeléctrica se realizarán varias actividades de manera paralela al diseño y evaluación de efectividad, como puede observarse en el cronograma. Además, los análisis que se realicen en esta fase se harán a partir de información secundaria, a excepción de la valoración económica que se espera desarrollar con información primaria. Los indicadores que se obtengan buscarán evidenciar la factibilidad, y la validación técnica y comercial, dando una explicación de la dinámica del producto en el entorno económico en que se encuentra.

Inicialmente, se realizará la descripción comercial para poder desarrollar la tecnología, identificando las restricciones y/o características comerciales que se tienen para explotarla. En el caso de la protección, se definirá el tipo de patente que se debe solicitar de acuerdo al tipo que mejor se adapte a las características específicas del producto según su grado de novedad, nivel inventivo y aplicación industrial (*i.e.* patente de invención, de modelo de utilidad o de diseño industrial). Además de esta solicitud, se realizará un registro INVIMA nuevo y uno de modificación que permitan comercializar la tecnología desarrollada. Así mismo, se adaptará la tecnología al plan de explotación comercial de la empresa, buscando ampliar el mercado actual. Para ello se analizarán los posibles clientes y canales del proceso, desde el usuario hasta el pagador de la prótesis. Dado que se pretende incluir el escaneo 3D dentro del nuevo proceso de manufactura, se debe explorar el mercado nacional por medio de diferentes aliados comerciales en las principales ciudades del país. Para esto se estudiarán las diferentes entidades haciendo uso de un estudio de mercado creado por la empresa Cuántica de la Incubadora de empresa CREAME.

Luego, se realizarán encuestas a las personas que directa e indirectamente se encuentran involucrados con la prótesis (e.g. EPS, ARL, hospitales, ortopédicas, amputados transradiales, entre otros) en la que expresarán en unidades monetarias el valor que estarían dispuestos a pagar por la nueva prótesis, además de obtener su opinión sobre el producto que se pretende comercializar, para capturar así su interés; esto nos permitirá hacer la valoración económica de la tecnología. Así mismo, se proyectarán los estados de resultados y flujo de caja de la tecnología para al menos los próximos 5 años con el fin de entender el desempeño y viabilidad económica con base en los ingresos y egresos relacionados con la producción y comercialización. Dentro de los indicadores financieros se evaluarán los indicadores operativos (i.e. margen bruto y margen operacional) y los indicadores estratégicos (i.e. margen EBITDA y ciclo de caja) para medir la evolución y compararlo con la industria, definiendo así la generación de valor económico de la tecnología. En este mismo sentido, y con base en la caja generada de la empresa, se aplicará el método de valoración de flujo de caja libre descontado, el cual permitirá medir con base en las inversiones que requiere el desarrollo de la tecnología, la tasa interna de retorno (TIR) que de obtiene comparándola con la de mercado y definiendo así la escalabilidad y sostenibilidad financiera en el tiempo. Esto nos permitirá establecer la capacidad que tiene la prótesis de generar recursos y flujo de caja. Adicionalmente, se comparará y se complementará con el tipo de protección intelectual que se seleccione, por medio de lo invertido tanto en efectivo como en especie, y así agregarlo a la valoración económica del flujo de caja descontado.

A continuación, se realizará el estudio de factibilidad técnica, económica y financiera del proyecto. Para la factibilidad técnica se comprobará la utilidad de la prótesis (esta actividad

está incluida en la fase anterior de la metodología) y el valor agregado que tiene con respecto a los otros productos que ofrece el mercado nacional, a partir del concepto técnico de los expertos en salud vinculados al proyecto. A nivel económico se evaluará que la prótesis se pueda vender en el entorno deseado (e.g. EPS, ARL, privados etc.), generando un impacto positivo en las dinámicas comerciales al permitir el retorno a su trabajo previo, o a uno similar, a las personas a las que les sea adaptadas este tipo de prótesis; o en el caso que puedan realizar actividades que sin la adaptación de esta prótesis no consideraban posibles. Una vez se tenga la validación de la disposición del mercado a pagar por la tecnología, se proyectará la generación de caja que resulta de los ingresos por la venta y los costos y gastos en que se debe incurrir, y adicionalmente se integrarán las necesidades de capital de trabajo y sus posibles fuentes de financiación. Esta mezcla, permitirá entender la capacidad de la tecnología de generar ventas suficientes para darle sostenibilidad a la empresa y el sentido económico de la tecnología para mantenerse en el tiempo y apalancar los crecimientos proyectados.

Para la validación técnica y pre-comercial de la nueva prótesis mioeléctrica, además de las actividades realizadas en la fase anterior de la metodología, se analizará la competencia y se evaluará si el precio del producto es competitivo en el mercado nacional; se identificarán los posibles compradores de la nueva tecnología (e.g. EPS, ARL, privados etc.) y sus volúmenes de compra; y se establecerá el modelo de negocio del producto. Para establecer el modelo de negocio se aplicará el modelo Canvas, donde a través de nueve cuadros se determinarán los segmentos importantes del modelo: problema, soluciones actuales, recursos clave, propuesta de valor, clientes, canales de clientes, relación con clientes, estructura de costos y estructura de ingresos. Así mismo, se propone realizar una prueba piloto de comercialización con la entidad ARL Sura, en la cual se analizará el canal desde el accidente de trabajo, la atención médica, la rehabilitación, la valoración, la evaluación por parte de Prótesis Avanzadas, la cotización del servicio, el diseño del mismo, la fabricación, la adaptación al usuario, el entrenamiento, la entrega oficial, y el cobro por el servicio. De esta manera se recorrerán todos los pasos importantes en un proceso de comercialización, con el fin de evidenciar oportunidades de mejora.

# **CRONOGRAMA**

| Antividados | | Meses | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Actividades | 1 | 3 | 5 | 7 | 9 | 11 | 13 | 15 | 17 | 19 | 21 | 23 | 25 | 27 | 29 | 31 | 33 | 35 |
| Diser | io conceptual | | | | | | | | | | | | | | | | | | |
| 1.1 (1) | Planteamiento del árbol de objetivos | | | | | | | | | | | | | | | | | | |
| 1.2 | Establecimiento de las funciones | | | | | | | | | | | | | | | | | | |
| 1.3 | Especificación de los requerimientos de diseño | | | | | | | | | | | | | | | | | | |
| 1.4 | Determinación de las características de las prótesis comparando los requerimientos con el punto de vista de los usuarios (grupo focal) | | | | | | | | | | | | | | | | | | |
| 1.5 | Generación de alternativas de diseño | | | | | | | | | | | | | | | | | | |
| 1.6<br>(6) | Evaluación de las alternativas de diseño (grupo focal) | | | | | | | | | | | | | | | | | | |
| | ENTREGABLES: Informe del diseño conceptual | | | | | | | | | | | | | | | | | | |
| Diser | no de materialización | | | | | | | | | | | | | | | | | | |
| 2.1 (7) | Estudio de normas y estándares | | | | | | | | | | | | | | | | | | |
| 2.2 | Ejecución de cálculos | | | | | | | | | | | | | | | | | | |
| 2.3 | Realización de experimentos | | | | | | | | | | | | | | | | | | |
| 2.4 | Definición de los bocetos detallados | | | | | | | | | | | | | | | | | | |
| 2.7 | Evaluación de cumplimiento de criterios técnicos | | | | | | | | | | | | | | | | | | |
| 2.8 | Evaluación de cumplimiento de criterios económicos | | | | | | | | | | | | | | | | | | |
| 2.9 | Generación de los archivos CAD preliminares para impresión 3D | | | | | | | | | | | | | | | | | | |
| 2.10 | Fabricación de prototipo preliminar | | | | | | | | | | | | | | | | | | |

| A (1.11.1 | | Meses | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Actividades | 1 | 3 | 5 | 7 | 9 | 11 | 13 | 15 | 17 | 19 | 23 | 25 | 27 | 29 | 31 | 33 | 35 |
| 2.11 | Redacción del primer informe de | | | | | | | | | | | | | | | | | |
| (15) | avance técnico y financiero | | | | | | | | | | | | | | | | | |
| | ENTREGABLES: Primer informe de | | | | | | | | | | | | | | | | | |
| | avance técnico y financiero, e informe del | | | | | | | | | | | | | | | | | |
| | diseño de materialización | | | | | | | | | | | | | | | | | |
| Diser | no de detalle | | | | | | | | | | | | | | | | | |
| 2.11 | Ejecución de pruebas de producción y | | | | | | | | | | | | | | | | | |
| (16) | desempeño | | | | | | | | | | | | | | | | | |
| 2.12 | Realización de cambios en el diseño de | | | | | | | | | | | | | | | | | |
| 2.12 | acuerdo a resultados de las pruebas | | | | | | | | | | | | | | | | | |
| 2.13 | Generación de los archivos CAD | | | | | | | | | | | | | | | | | |
| | definitivos para impresión 3D | | | | | | | | | | | | | | | | | |
| 2.14 | I I | | | | | | | | | | | | | | | | | |
| 2.15 | Redacción del manual de uso de la | | | | | | | | | | | | | | | | | |
| (20) | prótesis | | | | | | | | | | | | | | | | | |
| | ENTREGABLES: Archivos CAD, lista de | | | | | | | | | | | | | | | | | |
| | partes y manual de usuario | | | | | | | | | | | | | | | | | ı |
| | ación de efectividad | | | | | | | | 1 | 1 | T T | | | 1 | | ı | 1 | |
| 3.1 | Definición de protocolos para la evaluación | | | | | | | | | | | | | | | | | |
| (21) | pre-comercial del prototipo | | | | | | | | | | | | | | | | | |
| 3.2 | Fabricación de prototipos para pruebas | | | | | | | | | | | | | | | | | |
| 3.3 | Evaluación de efectividad (funcionalidad, | | | | | | | | | | | | | | | | | |
| 0.0 | desempeño, calidad de vida, satisfacción) | | | | | | | | | | | | | | | | | |
| 3.4 | Redacción del segundo informe de | | | | | | | | | | | | | | | | | |
| | avance técnico y financiero | | | | | | | | | | | | | | | | | |
| 3.5 | Análisis estadístico de los resultados | | | | | | | | | | | | | | | | | |
| 3.6 | Redacción del artículo | | | | | | | | | | | | | | | | | |
| (26) | | | | | | | | | | | | | | | | | | |
| | ENTREGABLES: Prototipos; resultados | | | | | | | | | | | | | | | | | |
| | de pruebas de modularidad, funcionalidad, | | | | | | | | | | | | | | | | | |
| | desempeño, calidad de vida y satisfacción; | | | | | | | | | | | | | | | | | |
| | archivos actualizados a partir del resultado | | | | | | | | | | | | | | | | | |

| Actividades | | Meses | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Actividades | | 3 | 5 | 7 | 9 | 11 | 13 | 15 | 17 | 19 | 21 | 23 | 25 | 27 | 29 | 31 | 33 | 35 |
| | de las pruebas; artículo sometido e informe final | | | | | | | | | | | | | | | | | | |
| Análi | sis financiero, económico y comercial | | | | | | , | | | , | | | | | | , | | | |
| 4.1<br>(27) | Selección del tipo de derechos de protección de propiedad intelectual y solicitud | | | | | | | | | | | | | | | | | | |
| 4.2 | Solicitud de registros INVIMA | | | | | | | | | | | | | | | | | | |
| 4.3 | Plan de explotación comercial | | | | | | | | | | | | | | | | | | |
| 4.4 | Realización de encuestas | | | | | | | | | | | | | | | | | | |
| 4.5 | Valoración económica de la tecnología | | | | | | | | | | | | | | | | | | |
| 4.6 | Definición de la escalabilidad y sostenibilidad financiera en el tiempo | | | | | | | | | | | | | | | | | | |
| 4.7 | Estudio de factibilidad técnica, económica y financiera | | | | | | | | | | | | | | | | | | |
| 4.8 | Análisis del modelo de negocio | | | | | | | | | | | | | | | | | | |
| 4.9 | Prueba piloto de comercialización | | | | | | | | | | | | | | | | | | |
| 4.10<br>(36) | Redacción de informe final técnico y financiero | | | | | | | | | | | | | | | | | | |
| | <b>ENTREGABLES:</b> Solicitud de derechos de protección de propiedad intelectual, certificados INVIMA, informe final técnico y financiero | | | | | | | | | | | | | | | | | | |

## **PRODUCTOS Y RESULTADOS ESPERADOS**

Este proyecto será la base de una ambiciosa línea de investigación en el diseño y evaluación de tecnologías médicas, que permitirá la colaboración entre los grupos GIBIC y Rehabilitación en Salud para hacer las veces de los departamentos de I+D de pequeñas y medianas empresas que produzcan y comercialicen dispositivos médicos. Al finalizar el proyecto se esperan los siguientes resultados:

## **Obligatorios**

- Primer informe de avance técnico y financiero, que incluya:
  - Informe del proceso de construcción del prototipo de la tecnología.
  - Solicitud de derechos de protección de propiedad intelectual.
  - Videos o fotografías del prototipo funcional de la tecnología.
  - Los avances en los protocolos para la evaluación pre-comercial el prototipo.
- Segundo informe de avance técnico y financiero, que incluya:
  - Registros y certificaciones que aplican según el tipo de tecnología desarrollada.
  - Protocolos para la evaluación pre-comercial del prototipo.
- Informe final técnico financiero, que incluya:
  - Plan para la explotación comercial de la tecnología.
  - Valoración económica de la tecnología expresada en términos monetarios.
  - Estudio de factibilidad técnica, económica y financiera el proyecto empresarial para explotación comercial de la tecnología.
  - Validación técnica y pre-comercial de la tecnología o sus productos y procesos derivados, incluyendo evidencias de acercamiento o comercialización con usuarios o clientes finales.

#### Además, se espera obtener los siguientes resultados:

- Una (1) patente solicitada sobre el diseño de la prótesis.
- Dos (2) artículo aceptados para publicación en revistas indexadas de clasificación A o B sobre el desarrollo y/o evaluación de efectividad de la nueva prótesis.
- Dos (2) trabajos aceptados para ponencias en eventos científicos nacionales o internacionales.
- Vinculación de un (1) estudiante de maestría de la Universidad de Antioquia.

# **POSIBLES EVALUADORES**

Juan Fernando Ramírez

Correo: <u>iframirp@unal.edu.co</u> Teléfono: 311 369 0444

Juan Pablo Valderrama

Correo: pablovalderrama@yahoo.com

Teléfono: 311 771 6353

Marcela Cristina Múnera Ramírez

Correo: marcela.munera@esculeaing.edu.co

# **BIBLIOGRAFÍA**

- [1] World Bank, «Discapacidad», World Bank, 03-abr-2019. [En línea]. Disponible en: http://www.bancomundial.org/es/topic/disability. [Accedido: 15-may-2019].
- [2] World Health Organization, «WHO | Disability and rehabilitation: WHO action plan 2006-2011», WHO. [En línea]. Disponible en: http://www.who.int/disabilities/publications/action\_plan/en/. [Accedido: 15-jun-2015].
- [3] Naciones Unidas Personas con Discapacidad, «Algunos datos sobre las personas con discapacidad | Disabilities ES», *Naciones Unidas*. [En línea]. Disponible en: https://www.un.org/development/desa/disabilities-es/algunos-datos-sobre-las-personas-con-discapacidad.html. [Accedido: 15-may-2019].
- [4] E. Cutillas Orgilés, «Distribución mundial de la población con discapacidades en relación con los patrones geográficos del desarrollo humano», *Doc. Anàlisi Geogràfica*, vol. 63, n.º 1, p. 29, ene. 2017.
- [5] Ministerio de Salud y Protección Social. Oficina de Promoción Social, «Sala situacional de las Personas con Discapacidad», jun-2018.
- [6] K. Ziegler-Graham, E. J. MacKenzie, P. L. Ephraim, T. G. Travison, y R. Brookmeyer, «Estimating the Prevalence of Limb Loss in the United States: 2005 to 2050», Arch. Phys. Med. Rehabil., vol. 89, n.º 3, pp. 422-429, mar. 2008.
- [7] C. Lake, «The Evolution of Upper Limb Prosthetic Socket Design», *JPO J. Prosthet. Orthot.*, vol. 20, n.º 3, p. 85, jul. 2008.
- [8] B. Rosenkrantz *et al.*, «Systems and methods for integrated robust orthotics and prosthetics hyper-customization», US20170285618A1, 05-oct-2017.
- [9] F. Cordella *et al.*, «Literature Review on Needs of Upper Limb Prosthesis Users», *Front. Neurosci.*, vol. 10, 2016.
- [10] J. M. Cancio, A. J. Ikeda, S. L. Barnicott, W. L. Childers, J. F. Alderete, y B. J. Goff, «Upper Extremity Amputation and Prosthetics Care Across the Active Duty Military and Veteran Populations», *Phys. Med. Rehabil. Clin. N. Am.*, vol. 30, n.º 1, pp. 73-87, feb. 2019.
- [11] C. Behrend, W. Reizner, J. A. Marchessault, y W. C. Hammert, «Update on Advances in Upper Extremity Prosthetics», *J. Hand Surg.*, vol. 36, n.º 10, pp. 1711-1717, oct. 2011.
- [12] DANE, «Estadísticas sobre Discapacidad», *Departamento Aadministrativo Nacional de Estadística*, 01-nov-2010. [En línea]. Disponible en: http://www.dane.gov.co/index.php/poblacion-y-demografia/discapacidad. [Accedido: 23-sep-2013].
- [13] Y. Ruiz, «Fabrilab: Imprimir calidad de vida en 3D», ELESPECTADOR.COM, 09-ago-2018. [En línea]. Disponible en: https://www.elespectador.com/noticias/bogota/fabrilab-imprimir-calidad-de-vida-en-3d-articulo-805185. [Accedido: 15-may-2019].
- [14] S. Watve, G. Dodd, R. MacDonald, y E. R. Stoppard, «Upper limb prosthetic rehabilitation», *Orthop. Trauma*, vol. 25, n.º 2, pp. 135-142, abr. 2011.
- [15] Y. Sang, X. Li, y Y. Luo, «Biomechanical design considerations for transradial prosthetic interface: A review», *Proc. Inst. Mech. Eng. [H]*, vol. 230, n.° 3, pp. 239-250, mar. 2016.
- [16] Congreso de Colombia, Ley de 1751 de 2015. 2015, p. 13.
- [17] Congreso de Colombia, Ley 1618 de 2013. 2013.
- [18] Congreso de Colombia, Ley 361 de 1997. 1997.
- [19] Congreso de Colombia, Ley 1295 de 1994. 1994.
- [20] Ministerio de Salud y Protección Socal, Ley 5857 de 2018. 2018.
- [21] K. Østlie, I. M. Lesjø, R. J. Franklin, B. Garfelt, O. H. Skjeldal, y P. Magnus, «Prosthesis rejection in acquired major upper-limb amputees: a population-based survey», *Disabil. Rehabil. Assist. Technol.*, vol. 7, n.º 4, pp. 294-303, jul. 2012.
- [22] E. Biddiss, D. Beaton, y T. Chau, «Consumer design priorities for upper limb prosthetics», *Disabil. Rehabil. Assist. Technol.*, vol. 2, n.º 6, pp. 346-357, ene. 2007.

- [23] A. Dabaghi-Richerand, F. Haces-García, y R. Capdevila-Leonori, «Prognostic factors of a satisfactory functional result in patients with unilateral amputations of the upper limb above the wrist that use an upper limb prosthesis», *Rev. Esp. Cir. Ortopédica Traumatol. Engl. Ed.*, vol. 59, n.º 5, pp. 343-347, sep. 2015.
- [24] L. Resnik, «Development and testing of new upper-limb prosthetic devices: Research designs for usability testing», *J. Rehabil. Res. Dev.*, vol. 48, n.º 6, p. 697, 2011.
- [25] T. Duong *et al.*, «Comparative Study of Functional Grasp and Efficiency Between a 3D-Printed and Commercial Myoelectric Transradial Prosthesis Using Able-Bodied Subjects: A Pilot Study», *JPO J. Prosthet. Orthot.*, vol. 29, n.º 3, p. 112, jul. 2017.
- [26] E. Biddiss y T. Chau, «The roles of predisposing characteristics, established need, and enabling resources on upper extremity prosthesis use and abandonment», *Disabil. Rehabil. Assist. Technol.*, vol. 2, n.º 2, pp. 71-84, mar. 2007.
- [27] E. Biddiss y T. Chau, «Upper-Limb Prosthetics: Critical Factors in Device Abandonment», *Am. J. Phys. Med. Rehabil.*, vol. 86, n.º 12, pp. 977-987, dic. 2007.
- [28] E. A. Biddiss y T. T. Chau, «Multivariate prediction of upper limb prosthesis acceptance or rejection», *Disabil. Rehabil. Assist. Technol.*, vol. 3, n.º 4, pp. 181-192, jul. 2008.
- [29] L. E. Pezzin, T. R. Dillingham, E. J. MacKenzie, P. Ephraim, y P. Rossbach, «Use and satisfaction with prosthetic limb devices and related services», *Arch. Phys. Med. Rehabil.*, vol. 85, n.º 5, pp. 723-729, may 2004.
- [30] L. E. Diment, M. S. Thompson, y J. H. Bergmann, «Three-dimensional printed upper-limb prostheses lack randomised controlled trials: A systematic review», *Prosthet. Orthot. Int.*, vol. 42, n.° 1, pp. 7-13, feb. 2018.
- [31] J. ten Kate, G. Smit, y P. Breedveld, «3D-printed upper limb prostheses: a review», *Disabil. Rehabil. Assist. Technol.*, vol. 12, n.° 3, pp. 300-314, abr. 2017.
- [32] I. Vujaklija y D. Farina, «3D printed upper limb prosthetics», *Expert Rev. Med. Devices*, vol. 15, n.° 7, pp. 505-512, jul. 2018.
- [33] S. B. Godfrey *et al.*, «The SoftHand Pro: Functional evaluation of a novel, flexible, and robust myoelectric prosthesis», *PLOS ONE*, vol. 13, n.º 10, p. e0205653, oct. 2018.
- [34] N. V. Iqbal, K. Subramaniam, y S. Asmi P., «Robust feature sets for contraction level invariant control of upper limb myoelectric prosthesis», *Biomed. Signal Process. Control*, vol. 51, pp. 90-96, may 2019.
- [35] M. Sartori, G. Durandau, S. Došen, y D. Farina, «Robust simultaneous myoelectric control of multiple degrees of freedom in wrist-hand prostheses by real-time neuromusculoskeletal modeling», *J. Neural Eng.*, vol. 15, n.º 6, p. 066026, oct. 2018.
- [36] M. Cognolato et al., «Hand Gesture Classification in Transradial Amputees Using the Myo Armband Classifier\* This work was partially supported by the Swiss National Science Foundation Sinergia project # 410160837 MeganePro.», en 2018 7th IEEE International Conference on Biomedical Robotics and Biomechatronics (Biorob), 2018, pp. 156-161.
- [37] L. Schmalfuss *et al.*, «A hybrid auricular control system: direct, simultaneous, and proportional myoelectric control of two degrees of freedom in prosthetic hands», *J. Neural Eng.*, vol. 15, n.º 5, p. 056028, ago. 2018.
- [38] A. Waris, I. K. Niazi, M. Jamil, K. Englehart, W. Jensen, y E. N. Kamavuako, «Multiday Evaluation of Techniques for EMG Based Classification of Hand Motions», *IEEE J. Biomed. Health Inform.*, pp. 1-1, 2018.
- [39] F. Clemente *et al.*, «Intraneural sensory feedback restores grip force control and motor coordination while using a prosthetic hand», *J. Neural Eng.*, vol. 16, n.° 2, p. 026034, feb. 2019.
- [40] E. D'Anna *et al.*, «A closed-loop hand prosthesis with simultaneous intraneural tactile and position feedback», *Sci. Robot.*, vol. 4, n.º 27, p. eaau8892, feb. 2019.
- [41] M. Ariyanto, R. Ismail, J. D. Setiawan, y E. P. Yuandi, «Anthropomorphic transradial myoelectric hand using tendon-spring mechanism», *TELKOMNIKA Telecommun. Comput. Electron. Control*, vol. 17, n.º 1, pp. 537-548, feb. 2019.

- [42] J. Fajardo, V. Ferman, A. Lemus, y E. Rohmer, «An Affordable open-source multifunctional upper-limb prosthesis with intrinsic actuation», en *2017 IEEE Workshop on Advanced Robotics and its Social Impacts (ARSO)*, 2017, pp. 1-6.
- [43] K. H. Lee, H. Bin, K. Kim, S. Y. Ahn, B.-O. Kim, y S.-K. Bok, «Hand Functions of Myoelectric and 3D-Printed Pressure-Sensored Prosthetics: A Comparative Study», *Ann. Rehabil. Med.*, vol. 41, n.º 5, pp. 875-880, oct. 2017.
- [44] S. A. Curline-Wandl y M. A. Ali, «Single channel myoelectric control of a 3D printed transradial prosthesis», *Cogent Eng.*, vol. 3, n.° 1, p. 1245541, dic. 2016.
- [45] J. Cabibihan, M. K. Abubasha, y N. Thakor, «A Method for 3-D Printing Patient-Specific Prosthetic Arms With High Accuracy Shape and Size», *IEEE Access*, vol. 6, pp. 25029-25039, 2018.
- [46] A. Nistler *et al.*, «Design and Development of a Myoelectric Transradial Prosthesis», Degree of Bachelor of Science, WORCESTER POLYTECHNIC INSTITUTE, 2017.
- [47] B. Stephens-Fripp, M. J. Walker, E. Goddard, y G. Alici, «A survey on what Australians with upper limb difference want in a prosthesis: justification for using soft robotics and additive manufacturing for customized prosthetic hands», *Disabil. Rehabil. Assist. Technol.*, vol. 0, n.° 0, pp. 1-8, mar. 2019.
- [48] P. Alvial *et al.*, «Quantitative functional evaluation of a 3D–printed silicone-embedded prosthesis for partial hand amputation: A case report», *J. Hand Ther.*, vol. 31, n.° 1, pp. 129-136, ene. 2018.
- [49] D. W. Sime, «Potential Application of Virtual Reality for Interface Customisation (and Pretraining) of Amputee Patients as Preparation for Prosthetic Use», en *Biomedical Visualisation: Volume 1*, P. M. Rea, Ed. Cham: Springer International Publishing, 2019, pp. 15-24.
- [50] Ottobock, «100 years of Ottobock Quality for life». [En línea]. Disponible en: https://www.ottobock.com/en/100-years-quality-for-life/. [Accedido: 31-may-2019].
- [51] Ottobock, «Michelangelo hand prosthesis». [En línea]. Disponible en: https://www.ottobock.com.au/prosthetics/upper-limb/solution-overview/axon-bus-prosthetic-system-with-michelangelo-hand/. [Accedido: 31-may-2019].
- [52] Ottobock, «MyoFacil prosthetic hand | Ottobock AU». [En línea]. Disponible en: https://www.ottobock.com.au/prosthetics/upper-limb/solution-overview/myofacil-prosthesis-system/. [Accedido: 31-may-2019].
- [53] K. Lorenz, «Electrohand 2000 for children», Ottobock. [En línea]. Disponible en: https://www.ottobockus.com/prosthetics/upper-limb-prosthetics/solutionoverview/electrohand-2000-for-children/. [Accedido: 31-may-2019].
- [54] Ottobock, «bebionic hand». [En línea]. Disponible en: https://www.ottobock.com.au/prosthetics/upper-limb/solution-overview/bebionic-hand/. [Accedido: 31-may-2019].
- [55] Touch Bionics, «Touch Bionics», *Touch Bionics*. [En línea]. Disponible en: http://touchbionics.com/. [Accedido: 15-may-2019].
- [56] Touch Bionics, «i-limb ultra», Touch Bionics. [En línea]. Disponible en: https://www.touchbionics.com/products/active-prostheses/i-limb-ultra. [Accedido: 31-may-2019].
- [57] Touch Bionics, «i-limb quantum», *Touch Bionics*. [En línea]. Disponible en: https://www.touchbionics.com/products/active-prostheses/i-limb-quantum. [Accedido: 31-may-2019].
- [58] Mobius Bionics, «LUKE Arm Detail Page», *Mobius Bionics*. [En línea]. Disponible en: http://www.mobiusbionics.com/luke-arm/. [Accedido: 31-may-2019].
- [59] G. Corley, «Handiii: A Sub \$300, 3D Printed, Smart-Phone Connected Bionic Arm (VIDEO) |», Medgadget, 24-mar-2015.
- [60] Innovation Match MX, «PROBIONICS S.A. DE C.V.» [En línea]. Disponible en: https://innovationmatchmx.com/probionics-s-a-de-c-v/. [Accedido: 31-may-2019].
- [61] Vincent Systems, «Prosthetics», *Vincent Systems*. [En línea]. Disponible en: https://vincentsystems.de/en/prosthetics/. [Accedido: 31-may-2019].

- [62] N. Cross, Engineering Design Methods: Strategies for Product Design, 3rd Edition, 3 edition. Chichester; New York: Wiley, 2000.
- [63] G. Pahl, W. Beitz, J. Feldhusen, K. H. Grote, K. Wallace, y L. T. M. Blessing, *Engineering Design: A Systematic Approach*, 3rd edition. London: Springer, 2006.
- [64] Jr. Byron Wm. Brown, «The Crossover Experiment for Clinical Trials», *Biometrics*, vol. 36, n.° 1, pp. 69-79, 1980.
- [65] T. A. Louis, P. W. Lavori, J. C. Bailar, y M. Polansky, «Crossover and Self-Controlled Designs in Clinical Research», *N. Engl. J. Med.*, vol. 310, n.° 1, pp. 24-31, ene. 1984.
- [66] W. Hill, P. Kyberd, L. Hermansson, S. Hubbard, Ø. Stavdahl, y S. Śwanson, «Upper Limb Prosthetic Outcome Measures (ULPOM): A working group and their findings», *JPO J. Prosthet. Orthot.*, vol. 21, pp. P69-P82, oct. 2009.
- [67] A. W. Heinemann, R. K. Bode, y C. O'Reilly, «Development and measurement properties of the Orthotics and Prosthetics Users' Survey (OPUS): A comprehensive set of clinical outcome instruments», *Prosthet. Orthot. Int.*, vol. 27, n.º 3, pp. 191-206, dic. 2003.
- [68] H. Burger, F. Franchignoni, A. W. Heinemann, S. Kotnik, y A. Giordano, «Validation of the orthotics and prosthetics user survey upper extremity functional status module in people with unilateral upper limb amputation», *J. Rehabil. Med.*, vol. 40, n.º 5, pp. 393-399. may 2008.
- [69] G. M. Jarl, A. W. Heinemann, y L. M. N. Hermansson, «Validity evidence for a modified version of the Orthotics and Prosthetics Users' Survey», *Disabil. Rehabil. Assist. Technol.*, vol. 7, n.º 6, pp. 469-478, nov. 2012.
- [70] L. Resnik, M. Borgia, B. Silver, y J. Cancio, «Systematic Review of Measures of Impairment and Activity Limitation for Persons With Upper Limb Trauma and Amputation», *Arch. Phys. Med. Rehabil.*, vol. 98, n.º 9, pp. 1863-1892.e14, 2017.
- [71] H. Y. N. Lindner, B. S. Nätterlund, y L. M. N. Hermansson, «Upper limb prosthetic outcome measures: review and content comparison based on International Classification of Functioning, Disability and Health», *Prosthet. Orthot. Int.*, vol. 34, n.° 2, pp. 109-128, jun. 2010.
- [72] C. for D. and R. Health, «Guidance for the Use of Bayesian Statistics in Medical Device Clinical Trials», *U.S. Food and Drug Administration*, 02-sep-2019. [En línea]. Disponible en: http://www.fda.gov/regulatory-information/search-fda-guidance-documents/guidance-use-bayesian-statistics-medical-device-clinical-trials. [Accedido: 31-may-2019].
- [73] Ministerio de Salud, Resolución Número 8430 de 1993, vol. 8430. 1993.
- [74] Department of Health, Education, and Welfare y National Commission for the Protection of Human Subjects of Biomedical and Behavioral Research, «The Belmont Report. Ethical principles and guidelines for the protection of human subjects of research», *J. Am. Coll. Dent.*, vol. 81, n.° 3, pp. 4-13, 2014.

## **NORMATIVIDAD**

En el Anexo 6 se puede observar el formato de consentimiento informado que será utilizado durante el desarrollo del proyecto.